

## Statistical Analysis Plan

NCT Number: NCT05084053

Title: A Phase 3 Study to Evaluate the Efficacy, Safety and Tolerability of TAK-771 for the Treatment of Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP) and Multifocal Motor Neuropathy (MMN) in Japanese Subjects

Study Number: TAK-771-3002

Document Version and Date: Version 3.0 / 17-Oct-2024

Certain information within this document has been redacted (ie, specific content is masked irreversibly from view) to protect either personally identifiable information or company confidential information.



### STATISTICAL ANALYSIS PLAN

Study Number: TAK-771-3002

licable terms of Use A Phase 3 Study to Evaluate the Efficacy, Safety and Tolerability of TAK-771 for the Treatment of Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP) and Multifocal Motor Neuropathy (MMN) in Japanese Subjects Local Use only and subject to

rotocol Version: Amendme
Protocol Date: 18-May-2022 Protocol Version: Amendment 2

# **REVISION HISTORY**

| Version | Approval Date | Primary Rationale for Revision |
|---|---|---|
| 1.0 | 19-Aug-2021 | [Not Applicable] |
| 2.0 | 10-Apr-2024 | Correction regarding Protocol revision (removal of unnecessary Endpoint descriptions). |
| | | Corrected to match Protocol description and italicized the same description in Protocol. |
| | | Added description clarifying the analysis. |
| | | Added the following section: |
| | | - 6.1.5 Study Information |
| | | Added the following section: - 6.1.5 Study Information - 6.3.3 CIDP history |
| | | - 6.3.4 MMN history |
| | | - 6.5 Prior/Concomitant Surgeries and Procedures |
| | | - 9.1.9 Missing Date Information for First Symptoms |
| | | <ul> <li>9.1.10 Missing Date Information for Diagnosis</li> </ul> |
| | | - 9.2 Definition of AESIs |
| | | Updated the description in following section: |
| | | - 1.1.2 Secondary Objectives |
| | | - 1.2.2.2 Efficacy |
| | | - 6.1 General Considerations |
| | | <ul> <li>6.1.4 Analysis Approach for Time-to-Event Variables</li> </ul> |
| | | - 6.2 Disposition of Subjects |
| | | - 6.3.2 Medical History |
| | | 6.4 Medication History and Concomitant Medications |
| | | - 6.4.1 Prior Medications |
| | | - 6.4.2 Concomitant Medications |
| | ,C | - 6.6.1.3 Supplementary Analysis |
| | -0( | - 6.6.2 Secondary Endpoints Analysis |
| | . (0 | - 6.6.3 Tertiary Endpoints Analysis |
| | CO, | - 6.7.1 Adverse Events |
| 1 de | a. For non-co | <ul> <li>6.7.1.1 Descriptive Analysis of Adverse Events per Infusion, per<br/>Subject, per Subject-Year</li> </ul> |
| 10 | Ť | - 6.7.2 Adverse Events of Special Interest |
| 13/ | | - 6.7.3 Clinical Laboratory Evaluations |
| 8 | | - 6.7.4 Vital Signs |
| 0, | | - 6.7.7 ADA Analysis |
| | | - 6.7.8 Extent of Exposure and Compliance |
| | | - 6.10 Other Analyses |
| | | - 8.0 CHANGES TO PROTOCOL PLANNED ANALYSES |
| | | - 9.1.3 Definition of Visit Windows |
| | | - 9.1.14 Character Values of Clinical Laboratory Variables |

| | 3.0 | 17-Oct-2024 | Added description of analysis sets for Epoch 2 analysis in section 5.0. |
|---|---|---|---|
| | | | Updated description mainly to clarify the analysis in Epoch 2. In addition, in each section, added the range of Epoch 2 data to be used in the 2nd interim analysis and final analysis. |
| | | | Updated the description in following section: |
| | | | 6.1: Added description of the start timing of each period and description of the serum IgG baseline. |
| | | | - 6.2: Added description to distinguish between the first 6 months in Epoch 2 and the subsequent periods. |
| | | | - 6.6.2-1: Added the item to be displayed in listing. |
| | | | - 6.6.3: Corrected a typo in an item in the PK analysis. (Changed "SD of the geometric mean" to "CV of the geometric mean") Regarding the analysis of data after day 120, a condition was added that non-relapse/worsen subjects would not be included in the analysis if there was only data for day 120 or less. |
| | | | - 6.7.7: Clarified definition of terms and analysis tables. |
| | | | - 6.7.8: Added classification of Epoch 2. |
| | | | - 6.10: Clarified the formula for each Epoch. |
| | | | Deleted the following section: - 6.6.2: "9. Change from pre-SC treatment baseline in R-ODS" in |
| | | | SAP v2.0 was deleted because it was a duplicate description with "6.6.2-3". |
| | | | Deleted unnecessary statements from section 8.0. Corrected table 6-8 in section 9.1.3. |
| | | | Added section 9.3. |
| | | CC | Added section 7.3. |
| | | Forhou | |
| Property | > | Ø. | |
| | te | , | |
| | 10 | | |
| | o'\ | | |
| les, | | | |
| ~0e, | | | |
| 0,0, | | | |

# TABLE OF CONTENTS

| 1.0 | OBJEC | CTIVES, ENDPOINTS AND ESTIMANDS | 9 |
|---|---|---|---|
| 1.1 | | jectives | |
| | 1.1.1 | Primary Objective | |
| | 1.1.2 | Secondary Objectives | 9 |
| | 1.1.3 | Tertiary Objectives | 9 |
| 1.2 | 2 Enc | dpoints | 9 |
| | 1.2.1 | Primary Objectives Secondary Objectives Tertiary Objectives dpoints Primary Endpoints Secondary Endpoints 2.1 Safety 2.2 Efficacy Tertiary Endpoints imands Y DESIGN STICAL HYPOTHESES AND DECISION RULES | 9 |
| | 1.2.2 | Secondary Endpoints | 9 |
| | 1.2 | .2.1 Safety | 9 |
| | 1.2 | .2.2 Efficacy | 10 |
| | 1.2.3 | Tertiary Endpoints | 10 |
| 1.3 | Est. | imands | 11 |
| 2.0 | STUD | Y DESIGN | 13 |
| 3.0 | STATI | STICAL HYPOTHESES AND DECISION RULES | 14 |
| 3.1 | Sta | tistical Decision Rules | 14 |
| 3.2 | 2 Sta | tistical Decision Rules | 14 |
| 3.3 | 8 Mu | Iltiplicity Adjustment | 14 |
| 4.0 | SAMP | LE-SIZE DETERMINATION | 14 |
| 5.0 | ANAL | YSIS SETSSTICAL ANALYSIS | 15 |
| 6.0 | | | |
| 6.1 | Gei | neral Considerations | |
| | 6.1.1 | Handling of Treatment Misallocations | |
| | 6.1.2 | Analysis Approach for Continuous Variables | |
| | 6.1.3 | Analysis Approach for Binary Variables | |
| | | Analysis Approach for Time-to-Event Variables | |
| | | Study Information | |
| | | sposition of Subjects | |
| 12 | 6.2.1 | Protocol deviations | |
| 4 | 6.2.2 | COVID-19 | |
| 6.3 | | mographic and Other Baseline Characteristics | |
| • | 6.3.1 | Demographics and Baseline Characteristics | |
| | 6.3.2 | Medical History | |
| | 6.3.3 | CIDP history | |
| | 634 | MMN history | 21 |

| 6.4 N | Iedication History and Concomitant Medications | 21 |
|---|---|---|
| 6.4.1 | Prior Medications | |
| 6.4.2 | Concomitant Medications | |
| 6.5 P | rior/Concomitant Surgeries and Procedures | |
| 651 | Prior Procedures | 23 |
| 6.5.2 | Concomitant Procedures | 23 |
| 6.6 E | fficacy Analysis | 23 |
| 6.6.1 | Concomitant Procedures fficacy Analysis Primary Endpoints Analysis 6.1.1 Derivation of Endpoints 6.1.2 Sensitivity Analysis | 23 |
| 6 | 6.1.1 Derivation of Endpoints | 23 |
| 6 | 6.1.2 Sensitivity Analysis | 24 |
| 6 | 6.1.3 Supplementary Analysis | 24 |
| 6.6.2 | Secondary Endpoints Analysis | 25 |
| 6 | 6.2.1 Sensitivity Analysis | 29 |
| 6 | 6.2.2 Supplementary analysis | 29 |
| 6.6.3 | 6.1.3 Supplementary Analysis | 29 |
| 6.7 S | afety Analysis | 31 |
| 6.7.1 | Adverse Events | 31 |
| 6 | 7.1.1 Descriptive Analysis of Adverse Events per Infusion, per Subject, p | ber |
| 6.7.2 | Subject-Year | |
| 6.7.2 | Adverse Events of Special Interest | |
| 6.7.3 | Clinical Laboratory Evaluations | |
| 6.7.4 | Vital Signs | 36 |
| 6.7.5 | ECG | |
| 6.7.6 | Clinically significant, treatment-emergent changes in physical exams | |
| 6.7.7 | ADA Analysis | |
| 6.7.8 | Extent of Exposure and Compliance | |
| | harmacokinetic, Pharmacodynamic, and Biomarker Analyses | |
| 6.8.1<br>6.8.2 | | |
| 10N | Pharmacodynamic Analysis | |
| 6.8.3 | Biomarker Analysis | 41 |
| | atient Reported Outcomes (PROs) and Health Care Utilization Endpoints nalysis | 41 |
| 6.9.1 | PRO Analysis | |
| 6.9.2 | Health Care Utilization Analysis | |
| | ther Analyses | |
| | iterim Analyses | |

| | ata Monitoring Committee/Internal Review Committee/ [Other Data Review ommittees] | 43 |
|---|---|---|
| | RENCES | |
| 8.0 CHAN | NGES TO PROTOCOL PLANNED ANALYSES | 45 |
| 9.0 APPE | NDIX | 46 |
| 9.1 Da | NDIXta Handling Conventions | 46 |
| 9.1.1 | General Data Reporting Conventions | 46 |
| 9.1.2 | Definition of Baseline | 46 |
| 9.1.3 | General Data Reporting Conventions Definition of Baseline Definition of Visit Windows Repeated or Unscheduled Assessments of Safety Parameters | 46 |
| 9.1.4 | Repeated or Unscheduled Assessments of Safety Parameters | 56 |
| 9.1.5 | Handling of Missing, Unused, and Spurious Data | 56 |
| 9.1.6 | Missing Date of Investigational Product | 56 |
| 9.1.7 | Missing Date of Investigational Product | 56 |
| 9.1 | (Therapies/Procedures) | 56 |
| 9.1 | 1.7.2 Incomplete Stop Date | 57 |
| 9.1.8 | Missing Date Information for Adverse Events | 58 |
| 9.1 | 1.8.1 Incomplete Start Date | 59 |
| 9.1 | 1.8.2 Incomplete Stop Date | 59 |
| 9.1.9 | Missing Date Information for First Symptoms | 59 |
| 9.1.10 | Missing Date Information for Diagnosis | 59 |
| 9.1.11 | Missing Severity Assessment for Adverse Events | 59 |
| 9.1.12 | Missing Seriousness of Adverse Events | 59 |
| 9.1.13 | Missing Relationship to Investigational Product for Adverse Events | 59 |
| 9.1.14 | Character Values of Clinical Laboratory Variables | 60 |
| 9.2 De | efinition of AESIs | 61 |
| | signment of R-ODS Centile Metric Scores | |
| 9.4 Ar | ålysis Software | 77 |
| 1 ste | | |
| LIST OF IN- | TEXT TABLES | |
| Table 1.a | Estimand Framework | 11 |
| Table 1.b | Estimand Framework | 12 |
| Table 2 | Criteria for Potentially Clinically Significant Vital Signs | 36 |
| Table 3 | Epoch 1 Analysis Windows for Efficacy Assessments in Subjects with SC Dosing Every 2 Weeks | 47 |

| | Table 4 | Epoch 1 Analysis Windows for Efficacy Assessments in Subjects with SC Dosing Every 3 Weeks | 48 |
|---|---|---|---|
| | Table 5 | Epoch 1 Analysis Windows for Efficacy Assessments in Subjects with SC Dosing Every 4 Weeks | 49 |
| | Table 6 | Epoch 2 Analysis windows for Efficacy Assessments (Dosing Every 2 | 50 |
| | Table 7 | Epoch 2 Analysis Windows for Efficacy Assessments (Dosing Every 3) | 52 |
| | Table 8 | Epoch 2 Analysis Windows for Efficacy Assessments (Dosing Every 4 Weeks) | 54 |
| | Table 9 | Weeks) | 61 |
| | Table 9.1 | Oedema of tongue, lips, face (angioedema) | 62 |
| | Table 9.2 | Anaphylaxis | 62 |
| | Table 9.3 | Persistent induration or nodule | 62 |
| | Table 9.4 | Excessive inflammation | 63 |
| | Table 9.5 | Adverse Events of Special Interest Oedema of tongue, lips, face (angioedema). Anaphylaxis Persistent induration or nodule Excessive inflammation Tissue necrosis/ulceration Dystrophic or fibrotic changes Pigmented skin changes | 63 |
| | Table 9.6 | Dystrophic or fibrotic changes | 64 |
| | Table 9.7 | Pigmented skin changes | 64 |
| | Table 9.8 | Rash | 64 |
| | Table 9.9 | Purpura | 65 |
| | Table 9.10 | Nephritis | 65 |
| | Table 9.11 | Arterial | 66 |
| | Table 9.12 | Venous | 70 |
| | Table 9.13 | Vessel unspecified/unknown | 72 |
| | Table 10 | R-ODS Score Conversion | 76 |
| Properti | orakedo | | |

### **ABBREVIATIONS**

ADL Activities of daily living

ΑE Adverse event AR Adverse reaction CI Confidence interval

CIDP Chronic Inflammatory Demyelinating Polyradiculoneuropathy

COVID-19 Coronavirus disease 2019 CRA Clinical research associate

CTMS Clinical Trial Management System

CVCoefficient of Variation

E1INT Epoch 1 interim E1W1 Epoch 1 Week 1

E<sub>0</sub>6M End-of-Epoch 2 (6 Months)

EoE1 End-of-Epoch 1

EoE2 End-of-Epoch 2 (continued)

**ECG** Electrocardiogram **FAS** Full analysis set

**GNDS** Guy's Neurological Disability Scale

Immunoglobulin G IgG

Inflammatory Neuropathy Cause and Treatment disability score **INCAT** 

ΙP **Investigation Product IVIG** Intravenous immunoglobulin

Medical Dictionary for Regulatory Activities MedDRA

MMN Multifocal Motor Neuropathy MRC Medical Research Council Potentially clinically significant **PCS** 

PK Pharmacokinetic Per-protocol set **PPS** 

Patient-reported outcomes **PRO** PT Preferred Term (MedDRA)

Rasch Built Overall Disability Scale R-ODS

Q1 1st quartile 3rd quartile

rHuPH20 Recombinant human hyaluronidase

SAE Serious adverse event SAP Statistical analysis plan SD Standard deviation SOC System Organ Class SYs Subject-years

TEAE Treatment-emergent adverse event

TIBC **Total Iron Binding Capacity** 

### 1.0 OBJECTIVES, ENDPOINTS AND ESTIMANDS

# 1.1 Objectives

## 1.1.1 Primary Objective

To evaluate the efficacy of TAK-771 in Epoch 1 as a maintenance therapy for Japanese patients with stable Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP) and Multifocal Motor Neuropathy (MMN) to prevent relapse or progression of motor function.

## 1.1.2 Secondary Objectives

- To assess the safety and tolerability of TAK-771 in Epoch 1 and Epoch 2 as a maintenance therapy for Japanese patients with CIDP and MMN
- To assess the efficacy of TAK-771 in Epoch 1 and Epoch 2

### 1.1.3 Tertiary Objectives

- To assess the serum trough levels of total immunoglobulin G (IgG)
- To assess the number of subjects using self-administration

### 1.2 Endpoints

### 1.2.1 Primary Endpoints

• Cohort 1 (CIDP)

Occurrence of relapse in Epoch 1 (worsening of functional disability defined as an increase of  $\geq 1$  point relative to the pre-SC treatment baseline score in adjusted Inflammatory Neuropathy Cause and Treatment (INCAT) disability score)

• Cohort 2 (MMN)

Change in maximum grip strength in the more affected hand in Epoch 1 (per baseline measurement point, investigators judge which of both hands is more affected)

### 1.2.2 Secondary Endpoints

### 1.2.2.1 Safety

- Cohort 1 (CIDP) and Cohort 2 (MMN)
  - Treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) regardless of causality
  - Causality of related SAEs and/or AEs
  - Serious and/or nonserious adverse reactions (ARs) plus suspected ARs\*
  - Treatment-emergent SAEs and/or AEs associated with infusions, regardless of causality

- Causality of related SAEs and/or AEs associated with infusions
- reins of Use AEs temporally associated with infusions (defined as AEs occurring during or within 72 hours after completion of an infusion)
- Serious and/or nonserious ARs plus suspected ARs associated with infusions
- Treatment-emergent systemic AEs associated with infusions
- Treatment-emergent local infusion site reactions associated with infusions
- Infusions for which the infusion rate was reduced and/or the infusion was interrupted or stopped due to intolerability and/or AEs
- Development positive titer ( $\geq 160$ ) binding antibodies, or develop neutralizing antibodies, to recombinant human hyaluronidase (rHuPH20)
- \* In the current study, an AR/suspected AR is defined as an AE that is considered by the investigator to be possibly or probably related to investigational product (IP) administration, or for which the causality is indeterminate or missing, or that begins during infusion of IP or within 72 hours following the end of IP infusion

### 1.2.2.2 **Efficacy**

- Cohort 1 (CIDP)
  - CIDP worsening in Epoch 1 (defined as  $a \ge 8$  kPa decrease in the hand grip strength in the more affected hand)  $OR \ge 4$  points decrease in Rasch-Built Overall Disability Scale (R-ODS) relative to the pre-SC treatment baseline score at 2 consecutive time points (at the time of withdrawal from the SC treatment period)
  - Time to relapse in Epoch 1 and Epoch 2
  - Change from pre-SC treatment baseline in R-ODS score in Epoch 1
  - Change from baseline in an average of handgrip strength of both hands in Epoch 1
- Cohort 2 (MMN)
  - Medical Research Council (MRC) sum score in Epoch 1
  - Gw's Neurological Disability Scale (GNDS) in upper limb and lower limb categories an Epoch 1

Change from baseline in an average of handgrip strength of both hands in Epoch 1

# **Tertiary Endpoints**

- Serum trough levels of total IgG
- Number of subjects received the study drug through self-administration

### 1.3 Estimands

Table 1.a Estimand Framework

| | ort 1 (CIDP) Attributes | | | |
|---|---|---|---|---|
| . , | Variable<br>(or Strategy for Ad<br>ent Population Endpoint) Intercurrent | - | Treatment | Definition |
| TAK-771 per subjects with a of relapse month will be adjusted to be equivalent to CIDP for subject's monthly approval intravenous (defined immunoglobulin (IVIG) dose. The appropriate AE, Significant protocol deviation, Voluntary withdrawal, Pregnancy, CIDP relapse, start the excluded medications or non-drug therapies, termination of TAK-771 administration by | er subjects with a of relapse be confirmed in Epoch 1 deviation, Volume withdrawal, Pregroom on the control of | subjects with a confirmed diagnosis of CIDP for approval (defined through appropriate inclusion/exclusion criteria) and who received TAK-771 at least once | TAK-771 per month will be adjusted to be equivalent to subject's monthly intravenous immunoglobulin (IVIG) dose. The number of infusion visits and site visits during the SC treatment period will vary across subjects depending on whether their infusion cycles | The primary estimand is the treatment effect of TAK-771 during Epoch 1 in targeted patient population. |

Table 1.b Estimand Framework

| Attributes Variable (or Strategy for Addressing Intercurrent Event Summary The IgG dose of Japanese Change in Early termination due to AE, The change in TAK-771 per subjects with a maximum Significant protocol deviation from the month will be confirmed grip Voluntary withdrawal, baseline to |
|---|
| is TAK-771 per subjects with a maximum Significant protocol deviation from |
| adjusted to be equivalent to Subject's approval affected monthly IVIG (defined hand in through dose. The number of infusion visits and site visits during the SC treatment period will vary across subjects depending on whether their infusion cycles are every 2, 3, or 4 weeks. Add. Add. Add. Pregnancy, CIDP relapses start the end of study visit the excluded medications or non-drug therapies. ElINT or EoEI) in maximum grip strength in the excluded medications or non-drug therapies. Elint or administration by investigator's determination and dealn are regarded as the Intercurrent Event. While on the end of study visit the end of study visit the excluded medications or non-drug therapies. ElINT or EoEI) in maximum grip strength in the excluded medications or non-drug therapies. Elint or end of the visits and it is excluded medications or non-drug therapies. Elint or end of the visits and it is excluded medications or non-drug therapies. Elint or end of the visits and it each or non-drug therapies. Elint or end of the visits and it each or non-drug therapies. Elint or end of the visits and it each or non-drug therapies. Elint or end of the visits and it each or non-drug therapies. Elint or end of the visits and it each or non-drug therapies. Elint or end or en |

are two treatment Epochs, with 2 cohorts of CIDP and MMN patients in this study. A schematic of the study design is shown in Figure 6-1 of the Protocol. Investigational product administration and site visit schedule are the same in Cohort 1 and Cohort 2.1 endpoint measurements differ.

This study will enroll subjects with a confirmed diagnosis of CIDP or MMN, who have remained on a stable dosing regimen (monthly equivalent dose of 0.4 to 2.4 g/kg BW with a dosing interval of 2 to 6 weeks) of IVIG therapy for at least 12 weeks prior to screening.

After informed consent is obtained, subjects will undergo screening and baseline procedures for the determination of eligibility and will continue to receive their own IVIG treatment at the same dose and dosing intervals prescribed prior to their entry into this study. No dosing adjustment of IVIG treatment is allowed except in cases of intolerability.

Eligible subjects will receive TAK-771 SC for a treatment period of 6 months in Epoch 1. The IgG dose of TAK-771 per month will be adjusted to be equivalent to subject's monthly IVIG dose. The number of infusion visits and site visits during the SC treatment period will vary across subjects depending on whether their infusion cycles are every 2, 3, or 4 weeks. If a subject with CIDP has met relapse criteria or a subject with MMN has been judged as being worsened by the investigator, the subject will be discontinued from the study treatment (See details in Section 7.4 of the Protocol). For safety and tolerability data, the sponsor set the minimum duration of Epoch 2 as 6 months. After the first 6 months of Epoch 2, if the subject is tolerating the drug well and voluntarily wishes to continue TAK-771 treatment, the subject can stay in the study until the commercial TAK-771 is available in each study site. After the first 6 months of Epoch 2, the investigator may adjust the dose of TAK-771 administration in every 3 months (See eails in property of Lakedai. For nondetails in Section 6.1.1 of the Protocol). Schedule of assessments is varied across the dosing interval (See the details in Appendix A of the Protocol).

### 3.0 STATISTICAL HYPOTHESES AND DECISION RULES

### 3.1 **Statistical Hypotheses**

ins of Use The primary objective of Epoch 1 is to evaluate the efficacy of TAK-771 as a maintenance therapy for CIDP to prevent relapse of neuromuscular disability and impairment. The following null hypothesis and alternative hypothesis will be tested as the estimated relapse rate in placebotreated patients of 57%:

- $H_0$ : Relapse rate  $\geq 57\%$
- H<sub>1</sub>: Relapse rate <57%

When the upper bound of exact 2-sided Clopper-Pearson 95% CI for the relapse rate will be below the threshold of 57%, H<sub>0</sub> will be rejected.

### 3.2

Not applicable.

### 3.3

Not applicable.

### 4.0

Cohort 1 (CIDP)

Adjustment

Adjust The latest meta-analysis (Lewis et al., 2020 [1]) reported that 43% of placebo-treated patients showed no deterioration in 5 placebo-controlled clinical studies, hence the estimated relapse rate in placebo-treated patients of 57%. The estimated relapse rate of Cohort 1 is 12% based on the average relapse rate in 2 clinical trials (13% in ICE study and 10% in the PATH extension study). As a result, the estimated sample size to show a statistically significant (at the 2.5% level) lower relapse rate than 57% with about 90% power would be 16 CIDP patients based on an assumed TAK-771 relapse rate of 12% and assuming a 15% dropout rate using a 95% two-sided Clopper-Pearson CI. This sample size was calculated based on simulation results from 100,000 trials.

# Cohort 2 (MMN)

The target number of MMN subjects was determined based on feasibility given the inclusion and exclusion criteria for this study. Multifocal motor neuropathy is less prevalent than CIDP. The annual number of MMN patients in Japan is estimated to be about 400 cases (Matsui, 2012 [2]).  $ar{F}$ ive subjects are scheduled to be included in this study. Since this study is planned to be conducted in parallel with the clinical trial of maintenance therapy with CIDP patients, an effort would be made to recruit additional subjects until enrollment period of CIDP study ends, even if enrollment of 5 subjects is completed.

### 5.0 ANALYSIS SETS

- Enrolled Set: The Enrolled Set will consist of all subjects who signed the informed consent and not screen failed.
- Epoch 2 Entered Subjects: The Epoch 2 Entered Subjects will consist of all subjects who completed End-of-Epoch 1 visit and received the first TAK-771 administration in Epoch 2.
- Full Analysis Set (FAS): All enrolled subjects who received TAK-771 at least once, this will be the efficacy analysis set.
  - Moreover, Epoch 2 Full Analysis Set contains subjects that meet the above criteria for Full Analysis Set in Epoch 2.
- Safety analysis set: All enrolled subjects who received TAK-771 administration at least once, this will be the safety analysis set.
  - Moreover, Epoch 2 Safety Analysis Set contains subjects that meet the above criteria for Safety Analysis Set in Epoch 2.
- Per Protocol Set (PPS): All enrolled subjects who received TAK-771 at least once, and had no major protocol deviations that may have a significant impact on the primary endpoint. Such protocol deviations will be determined prior to End of Epoch 1 through subject review meeting; PPS will be used for sensitivity and/or supportive analyses

Although efficacy data will be assessed for CIDP and MMN independently, safety will be assessed as integrated data from CIDP and MMN subjects. Data for the 2 Epochs will be presented separately.

### 6.0 STATISTICAL ANALYSIS

### 6.1 General Considerations

Start of Epoch 1, End of Epoch 1/Start of Epoch 2 and End of Epoch 2 are defined as follows:

- Start of Epoch 1 Epoch 1 Week 1 (E1W1)
- End of Epoch 1/Start of Epoch 2 (6 months): End-of-Epoch 1 (EoE1) assessments are to be conducted on the day of the first infusion in the Epoch 2 (6 months). This will mark the subjects' completion of the Epoch 1.
- End of Epoch 2 (6 months): End-of-Epoch 2 (6 months) (Eo6M) assessments are to be conducted on the day of the first infusion in the Epoch 2 (continued). This will mark the subjects' completion of the Epoch 2 (6 months).
- Start of Epoch 2 (continued): It is the first infusion in the Epoch 2 (continued).
- End of Epoch 2 (continued): EoE2 (continued) will be the date of discontinuation of study at EoE2 (continued).

The start datetime of Epoch 1, Epoch 2 (6 months) and Epoch 2 (continued) will be the datetime of the first infusion (the earlier of rHuPH20 or 10% IGI) of each period.

Two formal interim data analysis and a final analysis are planned for this study. (Section 6.11)

In the second interim analysis, the analysis will be performed with data at time points up to the "Epoch 2 (6 months)", and the final analysis will include data after "Epoch 2 (continued)".

Baseline value is defined as the pre-SC treatment baseline visit value, if non-missing. If missing then the Screening visit value will be used (if the screening visit value is non-missing). In other words, the latest available value before first SC treatment intake will be defined as baseline value.

For the lab results, baseline value is defined as the Epoch 1 Week1 (E1W1) visit value, if non-missing. If missing, then the Screening visit value will be used (if the screening visit value is non-missing).

For the serum IgG, baseline value is defined as the value collected at Baseline visit during Screening Period (according to Electronic Data Capture) even if this value is not the latest available value before first SC treatment intake.

All statistical analyses of relapse rates (primary and supplementary) will be analyzed using an exact 2-sided Clopper-Pearson 95% CI.

Unless otherwise specified, summaries of continuous variables (e.g., change from baseline) will display the following descriptive statistics: number of subjects (n), mean, median, standard deviation (SD), minimum, maximum. Means and medians and quartiles (if applicable) will be presented to 1 more decimal place than the recorded data. SDs will be presented to 2 more decimal places than the recorded data. BML averaged vital signs (e.g., diastolic/systolic blood pressure), and derived scores will be rounded to 1 decimal place for reporting.

Summaries of categorical and count variables will display the following: number of subjects (n), percentage (%) of subjects in the category, and number of outcomes/events/occurrences. Each summary containing a percentage will include a footnote stating the denominator that was used in calculating the percentage, unless the percentage is self-explanatory. Percentages will be presented to 1 more significant digit than the raw (actual) data. No percentages will be displayed if the number of subjects is 0.

Missing data due to the COVID-19 pandemic will not be handled any differently than missing data for other reasons.

## 6.1.1 Handling of Treatment Misallocations

Not applicable.

## 6.1.2 Analysis Approach for Continuous Variables

The corresponding analysis approach is described in Section 6.1.

### 6.1.3 Analysis Approach for Binary Variables

All statistical analyses of relapse rates (primary and supplementary) will be analyzed using an exact 2-sided Clopper-Pearson 95% CI.

### 6.1.4 **Analysis Approach for Time-to-Event Variables**

2. Ad subject to the applicable to the applicable by The corresponding analysis approach for "Time to discontinuation" is described in Section 6.2.

The corresponding analysis approach for "Time to relapse" is described in Section 6.6.2.

### 6.1.5 **Study Information**

Study Information will be presented and include the following categories:

- Date First Subject Signed Informed Consent Form
- Date of Data Cutoff
- MedDRA Dictionary Version
- WHO Drug Dictionary version
- SAS Version Used for Creating the Datasets

### 6.2 **Disposition of Subjects**

### Epoch 1

Disposition summaries will be presented for overall and by cohort and will include, but are not limited to, number and percentage of subjects in the following categories, where applicable:

- Screened
- Screen failed
- Primary reason for screen failure
- Enrolled
- Received IP
- Completed Epoch 1
- Discontinued study prematurely during Epoch 1
- Primary reason for premature discontinuation during Epoch 1
- Completed Epoch 1 but not entered Epoch 2
- Primary reason for completed Epoch 1 but not entered Epoch 2
- Entered Epoch 2

Subjects who discontinued study prematurely in Epoch 1 is defined as subjects who discontinued study during Epoch 1 and did not enter Epoch 2.

# Epoch 2

Disposition summaries will be presented for overall and by cohort and will include, but are not limited to, number and percentage of subjects in the following categories, where applicable:

- Entered Epoch 2
- Received IP in Epoch 2
- Completed Epoch 2 (6 months)
- Discontinued study prematurely during Epoch 2 (6 months)
- Primary reason for premature discontinuation in Epoch 2 (6 months)
- Entered Epoch 2 (continued)
- Discontinued study prematurely during Epoch 2 (continued)
- Primary reason for premature discontinuation in Epoch 2 (continued)
- Completed Epoch 2 (continued)
- Discontinued study prematurely during Epoch 2
- Primary reason for premature discontinuation in Epoch 2

The number of subjects by site will also be summarized for the Safety Analysis Set.

Subjects who discontinued study prematurely in Epoch 2 is defined as subjects who entered Epoch 2 and discontinued study prematurely. Subjects who received IP in Eo6M are defined as "Entered Epoch 2 (continued)".

Overall Discontinuation Rates will also be summarized for the Enrolled Set. An exact 2-sided Clopper-Pearson 95% CI will be used to show overall discontinuation rates. The following will be reported:

- number of subjects included in the analysis
- number (%) of subjects included in the analysis who discontinued
- estimated overall discontinuation rates and corresponding two-sided 95% CIs

Additionally, the following listings will be presented for each epoch:

- Disposition (Enrolled Set)
- Listing of all screen failures (i.e., subjects that have signed the informed consent, but did not pass screening)
- All subjects who prematurely discontinued the study will be listed for the Enrolled Set and the listing will include the primary reason for discontinuation. All AEs for subjects who prematurely discontinued will be presented.

As a further supplementary analysis, time to discontinuation for Epoch 1 and overall will be presented graphically. Time to discontinuation/completion will be calculated as:

date of Epoch 1 discontinuation (the last assessment) /completion—date of initial dose of IP in Epoch 1 + 1 (for Epoch 1)

and all subjects will be counted as having the event (i.e. no subjects will be censored). The corresponding cumulative incidence (1-survival) function will be estimated using Kaplan-Meier curves, where the vertical axis will represent the cumulative risk of discontinuation and the number of subjects at-risk over time will be displayed.

6.2.1 Protocol device:

Protocol deviations will be recorded in the IQVIA Clinical Trial Management System (CTMS) and will be classified as major or minor by the site staff, clinical research associate (CRA) and/or medical monitor. Such protocol deviations will be determined prior to database lock. Major/minor protocol deviations will be summarized by category, cohort and epoch for Safety Analysis Set. Protocol deviations will also be listed by subject and by site for the Safety Analysis Set.

Deviation categories will be included as part of the CTMS protocol deviations log and may Use only and include any of the following categories:

- Informed Consent Criteria
- Eligibility and Entry Criteria
- Concomitant Medication Criteria
- Laboratory Assessment Criteria
- Study Procedures Criteria
- Serious Adverse Event Criteria
- Randomization Criteria
- Visit Schedule Criteria
- Investigation Product (IP) Compliance
- Efficacy Criteria
- Administrative Criteria
- Source Document Criteria
- Regulatory or Ethics Approvals Criteria
- COVID-19
- Other Criteria

Additionally, for each epoch, a separate table and listing of protocol deviations related to the COVID-19 pandemic will be presented (Section 6.2.2). Protocol deviations which relate to the Epoch 1 Per-Protocol analysis set are described in Section 5.0.

A separate table and listing of protocol deviations related to the COVID-19 pandemic will be presented for each epoch. Missing data due to the COVID-19 pandemic will not be handled any differently than missing data for other reasons.

6.3 Demographic and Other Baseline Characteristics

6.3.1 Demographics and Baseline Characteristics

Descriptive summaries of demographic, baseline and screening characteristics separately for Epoch 1 and Epoch 2. Demographics and the country of the c

(years), age group ( $\leq 55, \geq 55$ ), sex, race and ethnicity. Characteristics at screening will include height (cm), weight (kg) and body mass index (kg/m<sup>2</sup>). Demographic, baseline and screening aly and subject only and subject of the last of the la characteristic summaries will be presented for the following analysis sets / epoch:

### Epoch 1

**FAS** 

overall and by cohort, in addition to:

Screen failures

### Epoch 2

FAS

overall and by cohort.

Listings of the demographic, baseline and screening characteristics will be provided for Enrolled Set.

### **Medical History** 6.3.2

Subject medical history will be coded using the Medical Dictionary for Regulatory Activities (MedDRA, version 24.0 or higher). Medical history is captured on the "MEDICAL HISTORY" eCRF form.

The number of subjects with any relevant past and current medical conditions/diseases will be tabulated by MedDRA system organ class (SOC) and preferred term (PT) for the Safety Analysis Set by each cohort. A subject will only be counted once within a particular SOC (or PT) even if he/she has multiple conditions/diseases in the same SOC (or PT). Presentation by SOC and PT will present SOC sorted alphabetically and PT within SOC by descending frequency.

Listings of medical history will be provided using the Safety Analysis Set.

### 6.3.3 CIDP history

Descriptive summaries of CIDP history at screening will be presented using the Safety Analysis Sets. This summary will include time since first CIDP symptoms (years), time since CIDP diagnosis (years), subject age at first diagnosis of CIDP.

Time Since First Symptoms will be calculated as follows:

Time Since First Symptoms (years) = ("Date of Informed Consent" – "Date of First Symptoms") / 365.25.

Time Since Diagnosis will be calculated as follows:

Time Since Diagnosis (years) = ("Date of Informed Consent" – "Date of Diagnosis") 365.25.

Subject Age at First Diagnosis of CIDP will be calculated as follows:

Subject Age at First Diagnosis of CIDP (years) = ("Date of Diagnosis" – "Date of Birth") / 365.25.

Listings of CIDP history will be presented using the Safety Analysis Sets.

### 6.3.4 MMN history

Descriptive summaries of MMN history at screening will be presented using the Safety Analysis Sets. This summary will include time since first MMN symptoms (years), time since MMN diagnosis (years), subject age at first diagnosis of MMN.

Time Since First Symptoms will be calculated as follows:

Time Since First Symptoms (years) = ("Date of Informed Consent" – "Date of First Symptoms") / 365.25.

Time Since Diagnosis will be calculated as follows:

Time Since Diagnosis (years) — "Date of Informed Consent" — "Date of Diagnosis") / 365.25.

Subject Age at First Diagnosis of MMN will be calculated as follows:

Subject Age at First Diagnosis of MMN (years) = ("Date of Diagnosis" – "Date of Birth") / 365.25.

Listings of MMN history will be presented using the Safety Analysis Sets.

### 6.4 Medication History and Concomitant Medications

Medication History and Concomitant Medications are captured on the "MEDICAL HISTORY", "MEDICATION HISTORY (IVIG)" and "CONCOMITANT MEDICATIONS" eCRF form.

Medication history and concomitant medications will be coded using the World Health Organization-Drug Dictionary (WHO-DD, Version 01MAR2021 or later).

For data presentation purposes, prior and concomitant medications are defined as follows ('time' implies date and time):

Prior medication

Any medication with start time prior to time of Epoch 1 IP administration.

### Concomitant medication

Any medication with start time at or after time of Epoch 1 IP administration, OR medications with start time prior to Epoch 1 IP administration but continuing at or after Epoch 1 IP administration.

Note that medications with start time prior to time of Epoch 1 IP administration and stop time after time of Epoch 1 IP administration will be counted as both prior and concomitant medications.

For medications with partial onset times, non-missing date parts will be used to determine if the medication is a concomitant or prior medication (see Section 9.1.7). If a determination cannot be made using the non-missing date parts as to when the medication occurred relative to the date of IP administration, then the medication will be classified as concomitant medication.

### **6.4.1** Prior Medications

Prior medications will be provided in subject data listing only using the Safety Analysis Set.

### 6.4.2 Concomitant Medications

Listings of concomitant medications will be presented using the Safety Analysis Set.

# 6.5 Prior/Concomitant Surgeries and Procedures

Prior/Concomitant Surgeries and Procedures (simply referred to as procedures) are captured on the "PRIOR SURGERY/PROCEDURE", "CONCOMITANT PROCEDURES" eCRF form.

For data presentation purposes, prior and concomitant procedures are defined as follows ('time' implies date and time):

• Prior procedure

Any procedures with start time prior to time of Epoch 1 IP administration.

Concomitant procedure

Any procedures with start time at or after time of Epoch 1 IP administration, OR procedures with start time prior to Epoch 1 IP administration but continuing at or after Epoch 1 IP administration.

Note that procedures with start time prior to time of Epoch 1 IP administration and stop time after time of Epoch 1 IP administration will be counted as both prior and concomitant procedures.

For procedures with partial onset times, non-missing date parts will be used to determine if the procedure is a concomitant or prior procedure (see Section 9.1.7). If a determination cannot be made using the non-missing date parts as to when the procedure occurred relative to the date of IP administration, then the procedure will be classified as concomitant procedure.

### 6.5.1

### 6.5.2

... subject data listing only using the Safety Analysis Set.

Concomitant Procedures

Concomitant procedures will be provided in subject data listing only using the Safety Analysis Set.

Efficacy Analysis

Primary Endnoise

### 6.6

### 6.6.1

The following analyses will be performed in Epoch 1. The same analyses as in Epoch1 will also be performed in Epoch 2 as an exploratory analysis.

### Cohort 1 (CIDP)

The primary analysis for Cohort 1 is based on occurrence of relapse (worsening of functional disability defined as an increase of ≥1 point relative to the pre-SC treatment baseline score in adjusted INCAT disability score).

An exact 2-sided Clopper-Pearson 95% CI will be used to show relapse rates, with missing outcomes imputed as no relapse. The following will be reported:

- number of subjects included in the analysis
- number (%) of subjects included in the analysis who relapsed
- estimated relapse rates and corresponding two-sided 95% CIs

The efficacy would be shown in the case that the upper bound of 95% CI for the relapse rate would be below the threshold of 57%.

### Cohort 2 (MMN)

The change from baseline in maximum grip strength will be presented for more affected hand using descriptive statistics and 2-sided 95% CI based on the FAS.

### 6.6.1.1 Derivation of Endpoints

### Cohort 1 (CIDP)

A relapse is defined as a worsening of functional disability such that there is an increase of  $\geq 1$ point relative to the pre-SC treatment baseline visit score in adjusted INCAT disability scores. For the primary analysis missing outcomes will be imputed as no relapse.

Adjusted INCAT disability scores are defined as follows:

Identical to INCAT score (using 10-point scale) except: INCAT upper extremity score that changed from 0 to 1 or from 1 to 0 will not be incorporated into overall INCAT score as it is not considered clinically meaningful.

The following adjusted scores are to be followed:

- An arm grade = 0 at pre-SC treatment baseline changing to arm grade = 1 at week z: adjusted scores at week z should be 0
- An arm grade = 1 at pre-SC treatment baseline changing to an arm grade = 0 at week x; adjusted scores at week x should be 1

At any time during the SC treatment period, unscheduled visit(s) may take place for a subject whose CIDP is worsening to assess whether the subject has an increase in the adjusted INCAT disability score by  $\geq 1$  point relative to the pre-SC treatment baseline score. INCAT assessment will be repeated during the pre-SC treatment baseline visit or early termination visit, as applicable, to confirm the subject's adjusted INCAT disability score has increased by  $\geq 1$  point relative to the pre-SC treatment baseline score, at which time the final determination of whether a subject has met relapse criteria will be made.

In the second interim analysis, the pre-SC treatment baseline data and the data in Epoch 2 (The first 6 months of Epoch 2) will be used to analyze the relapse in Epoch 2.

In the final analysis, the pre-SC treatment baseline data and the data in Epoch 2 (The first 6 months of Epoch 2 and Epoch 2 continued) will be used to analyze the relapse in Epoch 2.

### Cohort 2 (MMN)

Maximum grip strength is defined as the maximum of 3 measurements for grip strength in the more affected hand at each visit.

If a subject has no available post-dose data, that subject will be excluded from the analysis.

In the second interim analysis, the pre-SC treatment baseline data and the data in Epoch 2 (The first 6 months of Epoch 2) will be used to analyze the maximum grip strength in Epoch 2.

In the final analysis, the pre-SC treatment baseline data and the data in Epoch 2 (The first 6 months of Epoch 2 and Epoch 2 continued) will be used to analyze the maximum grip strength in Epoch 2.

6.6.1.2 Sensitivity Analysis

Not applicable.

6.6.1.3 Supplementary Analysis

The following supplementary analyses will be performed in Epoch 1.

## Cohort 1 (CIDP)

- 1. Changing the missing outcomes imputed as relapse.
- 2. Changing the strategy to address intercurrent events for the primary estimand from while on treatment to Principal stratum strategy where the stratum is restricted to subjects who did not have an intercurrent event.

- 3. Changing the population for the primary estimand from FAS to PPS.
- 4. Changing the strategy to address intercurrent events for the primary estimand from while on treatment to Composite variable strategy where all subjects are treated as "Relapse" subjects. except those who have no intercurrent events and are identified to be "No Relapse" at End of Epoch 1.

As for the primary analysis, an exact 2-sided Clopper-Pearson 95% CI will be used to show the applica relapse rates for these supplementary analyses.

### Cohort 2 (MMN)

Not applicable.

### 6.6.2 **Secondary Endpoints Analysis**

All secondary endpoints analyses will be based on the FAS population. The following analyses will be performed in Epoch 1. Analysis of time to relapse will also be performed for Epoch 2. The same analyses as in Epoch1 will also be performed in Epoch 2 as an exploratory analysis.

### Cohort 1 (CIDP)

## 1. Clinical worsening of CIDP

Clinical worsening of CIDP is defined as  $\geq 8$  kPa decrease in the hand grip strength in the more affected hand OR ≥4 points decrease in R-ODS relative to the pre-SC treatment baseline score at 2 consecutive time points (at the time of withdrawal from the SC treatment period). If 2 consecutive time points are across the different Epoch, it will be considered worsened in Epoch 1. This endpoint will be analyzed using an exact 2-sided Clopper-Pearson 95% CI, as described for the primary analysis (Section 6.6.1), with no imputation of missing values.

Additionally, the number and percentage of subjects meeting each component of worsening will be presented. A listing for worsening of functional disability will be presented for the FAS population. This Listing also displays the percentile-converted values according to the table 10 in Section 9.3.

Also perform the same analysis as above, with the following changes to the definition of Clinical worsening of CIDP.

Modified definition: Clinical worsening of CIDP is defined as ≥8 kPa decrease in the hand grip strength in the more affected hand OR  $\geq 4$  points decrease in R-ODS relative to the pre-SC treatment baseline score at 2 consecutive time points (at the time of withdrawal from the SC treatment period). If the final time point data corresponds to " $\geq 8$  kPa decrease in the hand grip strength in the more affected hand  $OR \ge 4$  points decrease in R-ODS relative to the pre-SC treatment baseline score ", also treat it as Clinical worsening of CIDP.

### 2. Time to relapse

Time to relapse is defined as time from the date of the first SC administration of TAK-771 to the date of relapse (where relapse is defined as in Section 6.6.1.1). For subjects who relapsed in Epoch 1, time to relapse will be calculated as:

date of relapse – date of initial dose of IP in Epoch 1 + 1.

Subjects who did not relapse in Epoch 1 will be censored with time to censoring calculated as:

date of Epoch 1 discontinuation/completion – date of initial dose of IP in Epoch 1 + 1.

In the analysis through Epoch1 and Epoch2, time to relapse will be calculated as:

date of relapse – date of initial dose of IP in Epoch 1 + 1.

Subjects who did not relapse in Epoch 1 and Epoch 2 will be censored with time to censoring calculated as:

In the second interim analysis: date of discontinuation/completion of Epoch 2 (The first 6 months of Epoch 2) – date of initial dose of IP in Epoch 1 + 1.

In the final analysis: last date of discontinuation/completion of Epoch 2 (The first 6 months of Epoch 2 or Epoch 2 continued) – date of initial dose of IP in Epoch 1 + 1.

The statistics presented will include but are not limited to:

- number of subjects included in the analysis
- number of subjects with event
- number of subjects censored
- percentiles (25th, 50th and 75th, if calculable), minimum and maximum for the cumulative incidence (1-survival) function, estimated using the Kaplan-Meier method

Additionally, the cumulative incidence (1-survival) function will be estimated using Kaplan-Meier curves, where the vertical axis will represent the cumulative risk of experiencing a relapse and the number of subjects at-risk over time will be displayed.

3. Change from pre-SC treatment baseline in R-ODS

The mean change in R-ODS score, activities of daily living (ADL), from pre-SC treatment baseline will be analyzed using descriptive statistics and 2-sided 95% CI (baseline is defined in Section 6.1). The last non-missing change will be used for subjects who discontinued early. Subjects without post-baseline R-ODS data will not be included in the analysis.

Descriptive statistics (n, mean, median, SD, 1st quartile(Q1), 3rd quartile(Q3), minimum, maximum) will be presented for R-ODS and change from pre-SC treatment baseline for each visit. Additionally, the statistics reported will include but are not limited to:

• estimated change from baseline and two-sided 95% CIs

An additional plot of mean change from pre-SC treatment baseline of R-ODS by timepoint will be presented for all timepoints (weeks), using the FAS population. A listing for R-ODS score and derived endpoints will also be presented for the FAS population.

The same analyses as in Epoch1 will also be performed in Epoch 2 as an exploratory analysis.

In the second interim analysis, the pre-SC treatment baseline data and the data in Epoch 2 (The first 6 months of Epoch 2) will be used to analyze the R-ODS in Epoch 2.

In the final analysis, the pre-SC treatment baseline data and the data in Epoch 2 (The first 6 months of Epoch 2 and Epoch 2 continued) will be used to analyze the R-ODS in Epoch 2.

4. Change from pre-SC treatment baseline in an average of handgrip strength of both hands

The secondary endpoints associated to Cohort 1 (CIDP), change from pre-SC treatment baseline in an average of handgrip strength of both hands, will be analyzed according to the methods for the primary endpoint for Cohort 2 (MMN) (defined in Section 6.6.1).

Average of grip strength is defined as an average of the two maximum values: maximum of the 3 measurements in the more affected hand and the maximum of the 3 measurements in the less affected hand at each visit.

The same analyses as in Epoch1 will also be performed in Epoch 2 as an exploratory analysis.

In the second interim analysis, the pre-SC treatment baseline data and the data in Epoch 2 (The first 6 months of Epoch 2) will be used to analyze the average of handgrip strength of both hands in Epoch 2.

In the final analysis, the pre-SC treatment baseline data and the data in Epoch 2 (The first 6 months of Epoch 2 and Epoch 2 continued) will be used to analyze the average of handgrip strength of both hands in Epoch 2.

5. Change from pre-SC treatment baseline in adjusted INCAT disability score

The exploratory analyses associated to Cohort 1 (CIDP), change from pre-SC treatment baseline in adjusted INCAT disability score, will be analyzed according to the methods for the primary secondary endpoint for Cohort 2 (MMN) (defined in Section 6.6.1). Subjects without post-baseline adjusted INCAT disability score data will not be included in the analysis.

Descriptive statistics (n, mean, median, SD, Q1, Q3, minimum, maximum) will be presented for adjusted INCAT disability score and change from pre-SC treatment baseline for each visit. Additionally, the statistics reported will include but are not limited to:

• estimated change from baseline and two-sided 95% CIs

An additional plot of mean change from pre-SC treatment baseline of adjusted INCAT disability score by timepoint will be presented for all timepoints (weeks), using the FAS population. A listing for adjusted INCAT disability score will also be presented for the FAS population.

The same analyses as in Epoch1 will also be performed in Epoch 2 as an exploratory analysis.

In the second interim analysis, the pre-SC treatment baseline data and the data in Epoch 2 (The first 6 months of Epoch 2) will be used to analyze the adjusted INCAT disability score in Epoch 2

In the final analysis, the pre-SC treatment baseline data and the data in Epoch 2 (The first 6 months of Epoch 2 and Epoch 2 continued) will be used to analyze the adjusted INCAT disability score in Epoch 2.

### Cohort 2 (MMN)

# 6. GNDS in upper limb and lower limb categories

The secondary endpoints associated to Cohort 2 (MMN), GNDS in upper limb and lower limb categories, will be descriptively analyzed as a binary variable indicating whether the score of a subject increased from baseline to the value at each post baseline, with no imputation of missing values. The following will be reported:

• number of subjects and number (%) of subjects with increased score from baseline in upper limb or lower limb categories

The same analyses as in Epoch1 will also be performed in Epoch 2 as an exploratory analysis.

In the second interim analysis, the pre-SC treatment baseline data and the data in Epoch 2 (The first 6 months of Epoch 2) will be used to analyze the GNDS in upper limb and lower limb categories in Epoch 2.

In the final analysis, the pre-SC treatment baseline data and the data in Epoch 2 (The first 6 months of Epoch 2 and Epoch 2 continued) will be used to analyze the GNDS in upper limb and lower limb categories in Epoch 2.

7. Change from pre-SC treatment baseline in MRC sum score

The secondary endpoints associated to Cohort 2 (MMN), change from pre-SC treatment baseline in MRC sum score will also be analyzed according to the methods for the primary endpoint for Cohort 2 (MMN) (defined in Section 6.6.1).

An additional plot of mean change from pre-SC treatment baseline of MRC sum score by timepoint will be presented for all timepoints (weeks), using the FAS population. A listing for MRC sum score will also be presented for the FAS population.

The same analyses as in Epoch1 will also be performed in Epoch 2 as an exploratory analysis.

In the second interim analysis, the pre-SC treatment baseline data and the data in Epoch 2 (The first 6 months of Epoch 2) will be used to analyze the GNDS in upper limb and lower limb categories in Epoch 2.

In the final analysis, the pre-SC treatment baseline data and the data in Epoch 2 (The first 6 months of Epoch 2 and Epoch 2 continued) will be used to analyze the GNDS in upper limb and lower limb categories in Epoch 2.

8. Change from pre-SC treatment baseline in an average of handgrip strength of both hands

The secondary endpoints associated to Cohort 2 (MMN), change from pre-SC treatment baseline in an average of handgrip strength of both hands, will be analyzed according to the methods for the primary endpoint for Cohort 2 (MMN) (defined in Section 6.6.1).

Average of grip strength of both hands is defined as an average of the two maximum values: maximum of the 3 measurements in the more affected hand and the maximum of the 3 measurements in the less affected hand at each visit.

The same analyses as in Epoch1 will also be performed in Epoch 2 as an exploratory analysis

In the second interim analysis, the pre-SC treatment baseline data and the data in Epoch 2 (The first 6 months of Epoch 2) will be used to analyze the average of handgrip strength of both hands in Epoch 2.

In the final analysis, the pre-SC treatment baseline data and the data in Epoch 2 (The first 6 months of Epoch 2 and Epoch 2 continued) will be used to analyze the average of handgrip strength of both hands in Epoch 2.

### 9. Change from pre-SC treatment baseline in GNDS

The secondary endpoints associated to Cohort 2 (MMN), change from pre-SC treatment baseline in GNDS, will be analyzed according to the methods for the primary endpoint for Cohort 2 (MMN)(defined in Section 6.6.1).

An additional plot of mean change from pre-SC treatment baseline of GNDS by timepoint will be presented for all timepoints (weeks), using the FAS population. A listing for GNDS score will also be presented for the FAS population.

The same analyses as in Epoch1 will also be performed in Epoch 2 as an exploratory analysis.

In the second interim analysis, the pre-SC treatment baseline data and the data in Epoch 2 (The first 6 months of Epoch 2) will be used to analyze the GNDS in Epoch 2.

In the final analysis, the pre-SC treatment baseline data and the data in Epoch 2 (The first 6 months of Epoch 2 and Epoch 2 continued) will be used to analyze the GNDS in Epoch 2.

### 6.6.2.1 Sensitivity Analysis

Not applicable.

# 6.6.2.2 Supplementary analysis

Not applicable.

# 6.6.3 Tertiary Endpoints Analysis

# 1. Serum trough levels of total IgG

Values below the lower limit of quantitation (LLOQ) will be considered as zero for descriptive statistics of serum trough concentrations of IgG. LLOQ for total serum trough levels of IgG is 1.72 g/L.

### Epoch 1

Analyses of serum trough concentrations of IgG will include subjects in the Epoch 1 Safety Analysis Set by cohort and overall. Serum trough concentrations of IgG will be summarized

using descriptive statistics (n, mean, SD, median, Q1, Q3, minimum, maximum, geometric mean, Coefficient of Variation (CV) of the geometric mean) and 2-sided 95% CI for mean and geometric mean by timepoints and each visit. Also, change from baseline will be tabulated. Plots of individual serum trough concentrations of IgG will be presented.

In addition, the relationship between serum IgG trough levels after day 120 (every 2-week dosing Epoch 1 W27/EoE1; every 3-week dosing Epoch 1 W26/EoE1, every 4-week dosing Epoch 1 W28/EoE1) or at the time of relapse status (relapse, no relapse for CIDP)/worsening status (MMN has been judged as being worsened by Investigator) will be assessed as an exploratory analysis. Serum trough concentrations of IgG will be summarized by relapse status (for CIDP)/ worsening status (MMN has been judged as being worsened by Investigator) and using descriptive statistics (n, mean, SD, median, Q1, Q3, minimum, maximum, geometric mean, CV of the geometric mean). Also, change from baseline will be tabulated. MMN worsening is defined as "Lack of Efficacy" or "Progressive Disease" of primary reason off study treatment. For subjects who relapsed/worsened in Epoch 1, the first recorded IgG level after relapse/worsen was selected for this analysis. For subjects who did not relapse/worsen in Epoch 1, the last recorded IgG level on treatment during Epoch 1 was selected for this analysis. For subjects who did not relapse/worsen and who had no IgG results after Day 120 are not included.

### Epoch 2

Analyses of serum trough concentrations of IgG for Epoch 2 will be presented for the Epoch 2 Safety Analysis Set by cohort and overall. Serum trough concentrations of IgG will be summarized using descriptive statistics (n, mean, SD, median, Q1, Q3, minimum, maximum, geometric mean, CV of the geometric mean) and 2-sided 95% CI for mean and geometric mean by timepoints and each visit. Also, change from baseline will be tabulated. Plots of individual serum trough concentrations of IgG will be presented.

In the second interim analysis, the pre-SC treatment baseline data and the data in Epoch 2 (The first 6 months of Epoch 2) will be used to analyze the serum trough concentrations of IgG in Epoch 2.

In the final analysis, the pre-SC treatment baseline data and the data in Epoch 2 (The first 6 months of Epoch 2 and Epoch 2 continued) will be used to analyze the serum trough concentrations of IgG in Epoch 2.

2. Number of subjects received the study drug through self-administration.

Number and percentage of subjects received the study drug through self-administration will be summarized by cohort and epoch for Safety Analysis Set.

For calculating number of subjects received the study drug, number of subjects received the 10% IGI will be used.

Subjects received the study drug through self-administration will also be listed for the Safety Analysis Set.

In the second interim analysis, the data in Epoch 2 (The first 6 months of Epoch 2) will be used to analyze the study drug through self-administration in Epoch 2.

In the final analysis, the pre-SC treatment baseline data and the data in Epoch 2 (The first 6 months of Epoch 2 and Epoch 2 continued) will be used to analyze the study drug through self-administration in Epoch 2.

### 6.7 Safety Analysis

Safety analyses will be mainly presented by cohort, Epoch and overall. Analyses for clinical laboratory evaluations and vital signs will be presented by cohort and visit. Continuous data (e.g., change from baseline in a lab parameter) will be summarized using the following descriptive statistics: number of subjects (n), mean, median, SD, minimum value, maximum value.

Categorical data (e.g., occurrence of AE) will be summarized in terms of number and percentage of subjects in the category, and, where applicable, number of outcomes/events/occurrences in the category.

For analysis of "adverse events", "adverse events of special interest" and "extent of exposure and compliance", the following data will be used.

In the second interim analysis, the data in Epoch 2 (The first 6 months of Epoch 2) will be used to analyze the safety analysis in Epoch 2.

In the final analysis, the data in Epoch 2 (The first 6 months of Epoch 2 and Epoch 2 continued) will be used to analyze the safety analysis in Epoch 2.

### 6.7.1 Adverse Events

All AEs will be coded using MedDRA (version 24.0 or higher) and then reported by MedDRA SOC and PT, and overall. Only TEAEs will be analyzed. Non-TEAEs will be listed only.

TEAEs are defined as adverse events that occurred during or after administration of the first dose of IP. TEAEs caused in Epoch 1 are defined as AEs that occurs on or after the start of study drug administration, and before the first dose of IP in Epoch 2. TEAEs caused in Epoch 2 are defined as AEs that began during or after administration of the first dose of IP in Epoch 2.

IP-related TEAE: Any TEAE that is recorded by the investigator as "Related" to IP will be considered IP-related AE, and any AE recorded as "Not Related" will be considered unrelated AE.

TEAEs temporally associated with infusion: These are defined as AEs occurring during or within 72 hours after completion of an infusion.

Any treatment-emergent adverse events which are answered "Yes" to Infusion-Related Reaction Flag is counted as an infusion associated TEAEs.

ARs/Suspected ARs: Adverse reactions (AR) plus suspected ARs are defined as TEAEs that are considered by the investigator to be related to IP administration, or for which the causality is indeterminate or missing, or that begins during infusion of IP or within 72 hours following the end of IP infusion.

For action taken with study treatment by TEAE, both action taken with rHuPH20 and action taken with 10% IGI are collected. If "Drug Withdrawn" is selected in either rHuPH20 or 10% IGI, then the TEAE will be treated as "TEAEs leading to prematurely discontinuation".

Any TEAE with the MedDRA High-Level Group Term (HLGT) = "Administration site reactions" will be considered a local TEAE. In addition, any TEAE with Injection Site Reaction Flag = "Yes" will be considered a local TEAE. All other TEAE's will be considered a systemic AE.

The following summaries will be provided (no statistical hypothesis testing is planned):

- Number and percentage of subjects with TEAEs by SOC and PT, and overall
- Number of TEAEs: SOC and PT, and overall

The following approaches will be used, where applicable:

- Overall summary: Any TEAE, TEAE related to IP, severe TEAE, severe TEAE related to IP, serious TEAE, serious TEAE related to IP, TEAE leading to early discontinuation, TEAE leading to death, TEAE temporally associated with infusion, infusion associated TEAE, local TEAE, systemic TEAE and ARs/Suspected ARs
  - Summaries by SOC and PT: In the summaries, SOC will be sorted alphabetically, and PT will be sorted within each SOC in descending frequency in the Total column (i.e., the Total column will be sorted in descending order after the sorting by SOC and PT)
  - Summaries by Maximum Severity: Subjects with multiple events in the same category are counted only once in that category, using the event with the greatest severity. Subjects with events in more than one category are counted once in each of those categories
  - If more than 1 TEAE occurs within the same PT for the same subject, then the subject will be counted only once for that PT using the most severe and most related occurrence for the summarization by severity and by relationship to IP. For example, if a subject experienced a mild headache not related to the IP, and a moderate headache related to IP, then the subject will be counted once for headache using the moderate headache related to IP
  - In AE incidence summaries, subjects with multiple events in the same category will be counted only once in the AE category. Subjects with events in more than one category will be counted once in each of the categories
  - In AE count summaries, multiple occurrences of the same AE will be counted multiple times
  - Note that, in addition to standard AE listings, the following subject data listing will be provided per regulatory request: Subjects who prematurely discontinued from the study, and all their treatment-emergent adverse events. The listing will be based on the Enrolled Set and display demographics, first and last dose dates (if known),

6.7.1.1 Descriptive Analysis of Adverse Events per Infusion, per Subject, per Subject-Year

The following summaries will be provided for Epoch 1 and overall (no statistical hypothesis testing is planned):

• Number of TEAT

- Number of TEAEs per infusion, by SOC and PT
- Number of TEAEs per subject, by SOC and PT
- Number of TEAEs per 1000 subject-years, by SOC and PT

AEs per 1000 subject-years summary adjusts for differences in subjects' durations in the study and differential dropout rates between treatment groups.

For number of AEs, multiple occurrences of the same AE in the same subject will be counted multiple times.

Number of AEs and AEs per 1000 subject-years (SYs) will be provided for all AEs (if analyzable), by SOC and PT.

The following calculations apply, where applicable:

- AEs per infusion = number of AEs / total number of infusions administered of 10% IGI to subjects in the analysis set ②
- AE per subject = number of AEs / total number of subjects in the analysis set
- AEs per 1000 SYs in Epoch  $1 = 1000 \times (\text{Total Number of AEs in Epoch 1 for all})$ subjects / Total SYs in Epoch 1)
- Total SYs in Epoch will be calculated by summing subjects' durations in Epoch through the end of Epoch. Each subject's duration will be calculated as: (last date of Epoch – date of initial dose of IP in the Epoch + 1) / 365.25. If the subject's last date in the Epoch is missing, then the date of last dose of IP will be used if available

The following AEs will be summarized per infusion, subject, and subject year:

- Any TEAE
  - Serious TEAEs
- **IP-Related TEAEs**
- IP-Related Serious/Non-Serious TEAEs
- TEAEs temporally associated with infusion
- Local/Systemic TEAEs
- IP-Related Local/Systemic TEAEs
- IP-Related Serious Local/Systemic TEAEs

- TEAEs That Occurred During or Within 72 Hours Post-Infusion
- ARs/Suspected ARs
- ARs/Suspected ARs temporally associated with infusion

### **6.7.2** Adverse Events of Special Interest

AEs of special interest will be coded using the MedDRA (version 24.0 or higher) and then reported by MedDRA PT, and overall.

Adverse events of special interest (source: Section 9.1.9.10 of the study protocol) include Oedema of tongue, lips, face (angioedema)
Anaphylaxis
Stevens-Johnson syndroma
Erythema the followings (see Section 9.2 for details of definitions):

- Allergic reactions

  - Erythema multiforme
  - Toxic epidermal necrolysis
- Immune complex mediated reactions Local
  - Induration/nodule at the site of administration that persists for more than 48 hours
  - Excessive inflammation at the site of administration severe redness, heat, swelling, and/or pain
  - Tissue necrosis/ulceration at the site of administration
  - Dystrophic or fibrotic changes at the site of administration
  - Pigmented skin changes at the site of drug administration
- Immune complex mediated reactions Systemic
  - Arthritis
  - Vasculitis (purpuric rash)
  - Glomerulonephritis hematuria, red cell casts in urine, progressive renal dysfunction
- Thrombotic and Embolic Events
  - Arterial (Embolic and thrombotic events, arterial 20000082 (SMQ))

- Venous (Embolic and thrombotic events, venous 20000084 (SMQ))
- Vessel unspecified/unknown (Embolic and thrombotic events, vessel type unspecified and mixed arterial and venous - 20000083 (SMQ)).

The following special interest AEs will be summarized:

- Any TEAE of special interest
- TEAEs of special interest by Antibody Status (subject having elevated anti-rHuPH20 antibody titers or not).

# 6.7.3 Clinical Laboratory Evaluations

Clinical laboratories are not explicitly stated in the study protocol as endpoints but are included in this SAP for further assessment of the safety profile. Raw (actual) clinical laboratory values (in SI units) and changes in raw values from baseline at each post-baseline assessment time point will be summarized as continuous variables. Shift from baseline to each assessment time point will be provided for categorical variables. Results will be tabulated. The following laboratory variables/parameters will be summarized, and the data will be listed in the subject data listing, as indicated. Other than following Lab parameters will be listed only.

| Hematology | The hematology panel will consist of hemoglobin, hematocrit, erythrocytes (i.e., red blood cell count), and leukocytes (i.e., [WBC]) with differential (i.e., basophils, eosinophils, lymphocytes, monocytes, neutrophils) and platelet counts, as well as absolute neutrophil count. | Summary and Listing |
|---|---|---|
| Clinical<br>Chemistry | The clinical chemistry panel will consist of sodium, potassium, chloride, bicarbonate, protein, albumin, ALT, serum total bilirubin, AST, ALP, LDH, BUN, serum creatinine, creatinine phosphokinase, glucose, haptoglobin, and lipase | Summary and Listing |
| Hemolytic Panel | The hemolytic panel includes Hgb, LDH, serum haptoglobin, plasma-free (unbound) Hgb, serum direct anti-globulin (direct Coombs) test, reticulocyte count, and urine hemosiderin. | Listing only |
| Hemoglobin A1C | HbA1c | Listing only |
| Serum Iron,<br>Ferritin, and Total<br>Iron Binding<br>Capacity (TIBC) | Serum iron, ferritin, and TIBC | Listing only |
| Urinalysis | Color, specific gravity, pH, protein, glucose, ketones, bilirubin, urobilinogen, blood, nitrite, and leukocyte esterase and a microscopic examination | Listing only |
| Pregnancy Test | Pregnancy tests for female subjects of childbearing potential | Listing only |
Summaries of shift from baseline (shift tables) will be produced for each parameter that has a reference range, using the categories: low (below the lower limit of the reference range), normal (within the reference range) and high (above the upper limit of the reference range).

In addition, shift from baseline summaries will be produced by toxicity Grade. Summaries will display number and percent of subjects whose laboratory values were assessed as Grade < 3, Grade 3, Grade 4, or missing at the pre-SC baseline, and at the post-baseline maximum Grade.

Laboratory parameters will be summarized tabularly and/or graphically using spaghetti-plots or scatterplots as follows: spaghetti-plots of clinical chemistry values by parameter and visit; scatterplots of ALT, AST, and bilirubin post-baseline versus baseline comparisons to normal range limits by parameter and visit; spaghetti-plots of hematology values by parameter and visit.

The following will be provided in subject data listings.

- Hematology values for subjects who met toxicity Grade ≥ 3 criteria for any hematology parameter
- Clinical Chemistry values for subjects who met toxicity Grade ≥ 3 criteria for any clinical chemistry parameter
- Hemolytic parameters panel for subjects who showed a reduction in Hgb level of 1g/dL or more at any time after the first full dose of IP treatment during the epoch

## 6.7.4 Vital Signs

Vital signs endpoints are not explicitly mentioned in the study protocol as endpoints but are included in this SAP to further assess the safety. Raw (actual) values for vital signs and their changes from baseline at each post-baseline assessment time point will be summarized by visit. Vital signs will also be summarized both graphically (spaghetti-plots).

A vital sign value will be considered potentially clinically significant (PCS) if it meets both the observed value criteria and the change from baseline criteria listed in Table 2. Number and percentage of subjects with PCS post-baseline values will be tabulated. Percentages will be calculated relative to the number of subjects with baseline and at least 1 post-baseline assessment. The numerator is the total number of subjects with at least 1 PCS post-baseline vital sign value in the specified period.

Table 2 Criteria for Potentially Clinically Significant Vital Signs

| Vital Sign Parameter | Flag | Criteria <sup>a</sup> | |
|---|---|---|---|
| 8 | | Observed Post-Baseline Value | Change from Baseline |
| Systolic blood pressure | High | ≥ 180 | Increase of $\geq 20$ |
| (mmHg) | Low | ≤ 90 | Decrease of $\geq 20$ |
| Diastolic blood pressure | High | ≥ 105 | Increase of $\geq 15$ |
| (mmHg) | Low | ≤ 50 | Decrease of $\geq 15$ |
| Pulse rate | High | ≥ 120 | Increase of $\geq 15$ |
| (beats per minute) | Low | ≤ 50 | Decrease of ≥ 15 |

| Weight (kg) | High | - | Increase of ≥ 7% |
|-------------|------|---|------------------------|
| | Low | - | Decrease of $\geq 7\%$ |

<sup>&</sup>lt;sup>a</sup> A post-baseline value is considered as a PCS value if it meets both criteria for observed value and change from baseline.

#### 6.7.5 **ECG**

Electrocardiogram (ECG) data (overall interpretation) will be provided in subject listing only. Note that clinically significant, treatment-emergent changes in ECGs will be recorded in the study database as AEs.

#### Clinically significant, treatment-emergent changes in physical exams 6.7.6

A star and sent-emergence of takeda. For non-commercial use of takeda. For non-commercial use of takeda. Clinically significant, treatment-emergent changes in physical exams data will be listed in the subject listing only. Note that clinically significant, treatment-emergent changes in physical

## 6.7.7

The immunogenicity endpoints corresponding to the immunology safety objective include:

- e immunogenicity endpoints corresponding to the immunology safety objective include:

  Anti-rHuPH20 antibody (binding and/or neutralizing antibodies to rHuPH20), specifically subjects with:

  High-binding antibodies

  Low-binding antibodies

  Abnormal or increased anti-rHuPH20 antibody titer

  Elevated anti-rHuPH20 antibodies

  Neutralizing antibodies measured

  Positive neutralizing antibodies

  Negative neutralizing antibodies

  i-rHuPH20 antibody titer ≥ 1:160" means "Positive hebinding antibodies" ""

"Anti-rHuPH20 antibody titer ≥ 1:160" means "Positive titers (≥ 1:160)" and is described as "High-binding antibodies". "Titer < 1:160" is described as "Low-binding antibodies".

High-binding antibodies at any time: Number of subjects who had at least one anti-rHuPH20 antibody titer  $\geq 1:160$  during treatment.

High-binding antibodies at specific visit: Number of subjects who had anti-rHuPH20 antibody titer  $\geq 1:160$  at the specific visit.

Low-binding antibodies at any time: Number of subjects with anti-rHuPH20 antibody titer < 1:160 for all data during treatment.

Low-binding antibodies at specific visit: Number of subjects who had anti-rHuPH20 antibody titer <1:160 at the specific visit.

A subject is defined as having (1) abnormal or (2) increased from baseline if the subject has (1) anti-rHuPH20 antibody titer of  $\geq 1:160$  or (2) if anti-rHuPH20 antibody titer is higher than the greater of  $\geq 1:160$  of the value at baseline.

A subject is defined as having elevated anti-rHuPH20 antibody titers if the subject has two consecutive anti-rHuPH20 antibody titers of  $\geq 1:160$  which are elevated from the subject's baseline titers.

Antibody titers may be reported as direct titers (positive integers) or as the inverse of the amount of diluent that is required to abolish a positive test result. Subjects who have two consecutive anti-rHuPH20 antibody titers of > 1:160 which are elevated from the subject's baseline titers will be classified as experiencing treatment-emergent development of anti-rHuPH20 antibodies at the first of the two time points.

Anti-rHuPH20 antibody development will be summarized (number of subjects (n), percentage (%) of subjects by category: elevated, neutralizing antibody measured, positive neutralizing antibodies, negative neutralizing antibodies, high-binding, low binding) by visit.

reins of Use All treatment-emergent AEs and related AEs in subjects with "anti-rHuPH20 antibody titers ≥ 1:160" will be presented in a subject data listing. For subjects with/without "\geq 1:160 or increased from baseline in anti-rHuPH20 antibody titer", with "elevated titers", and without "antirHuPH20 antibody titers ≥ 1:160", all treatment-emergent AEs will be presented.

Additionally, AEs experienced by each of the titer groups will be summarized:

- Subjects with positive anti-rHuPH20 antibody titers (≥ 1:160)
  - All AEs and related AEs reported before the first positive anti-rHuPH20 antibody titers (>1:160) confirmation
  - All AEs and related AEs reported after the first positive anti-rHuPH20 antibody titers (≥ 1:160) confirmation
- Subjects with any treatment emergent abnormal titer ( $\geq 1:160$ ) or increased from baseline in anti-rHuPH20 antibody titer
  - All AEs and related AEs reported before any  $\geq 1:160$  or increased from baseline
  - All AEs and related AEs reported after any  $\geq 1:160$  or increased from baseline
- AEs for subjects without any treatment emergent  $\geq 1.160$
- AEs for subjects with elevated titers.

For TEAEs and IP-related TEAEs in subjects with "anti-rHuPH20 antibody titers ≥ 1:160", summarizes by SOC and PT (see section 6.74) and per Infusion, per Subject, per Subject-Year (see section 6.7.1.1).

For TEAEs in subjects with "\ge 1:160 or increased from baseline in anti-rHuPH20 antibody titer", with "elevated titers", and without "anti-rHuPH20 antibody titers ≥ 1:160", summarizes by SOC and PT and per Infusion, per Subject, per Subject-Year.

If at least 5 subjects have elevated titers, then the descriptive analysis will be conducted to assess if there is any evidence of relationship between anti-rHuPH20 antibody titer (elevated, not elevated) and the occurrence of AEs of interest. The occurrence of AEs of interest will be summarized by anti-rHuPH20 antibody titer.

In addition, the analysis of any treatment emergent abnormal titer or increased from baseline in anti-rHuPH20 antibody titer will be performed to assess if there is any evidence of relationship between anti-rHuPH20 antibody titer (elevated, not elevated) and the occurrence of AEs.

Immunology related data after IP administration will also be listed.

#### 6.7.8 **Extent of Exposure and Compliance**

Exposure to IP and compliance will be summarized separately for the Epoch 1 and Epoch 2 Safety Analysis Set. Each study drug (10% IGI, rHuPH20) will be summarized separately.

The following will be presented descriptively:

number of infusions which were interrupted/stopped/dose reduced or rate reduced

- number of infusions excluding interrupted/stopped/dose reduced or rate reduced
- number of infusions for which the infusion rate was reduced and/or the infusion was interrupted or stopped and/or dose reduced due to intolerability and/or AEs
- treatment duration (months, as defined below).

Infusion compliance is calculated as the total number of applied infusions of each study drug (10% IGI, rHuPH20) including completed, interrupted, and stopped infusions, divided by the number of expected infusions, multiplied by 100. The number of expected infusions is based on the actual number of visits. Actual number of visits means the visit up to the data cut-off or end of treatment during the epoch.

Descriptive statistics (n, mean, SD, minimum, median, and maximum) or number of subjects and percentage, as applicable, will be presented by dosing regimen, cohort and overall.

Exposure is defined as the total duration of treatment with IP (in days), calculated as:

date of last dose of IP – date of initial dose of IP + 1.

For calculating duration of treatment with IP, date of dose of 10% IGI will be used.

Treatment duration will be summarized both as a continuous variable and using the following categories:

- <1 month
- 1 <3 months
- 3 < 6 months
- 6 <12 months
- 12 <18 months
- 18 <24 months
- $\geq$ 24 months
- $\geq 1$  month
- >3 months
- $\geq 6$  months
- $\geq$ 12 months
- $\geq$ 24 months

And Summary of IP Administration will be tabulated.

The following will be presented descriptively:

Total Number of Infusions Administered

- Number of Infusion Sites on the Body Per Infusion (1, 2, 3)
- Actual Infusion Volume (mL)
- Maximum Infusion Rate/ Site (mL/hr)
- Study Treatment Administration Performed (Study Subject, Investigator/Study Physician, Study Nurse, Caregiver)

Additionally, monthly dose equivalent and duration of infusion per dose of 10% IGI will be presented in Epoch 1.

Full dose is defined as the dose that is achieved after ramp-up and occurs at Epoch 1 Week 3 (Every 2 Weeks Regimen), Epoch 1 Week 5 (Every 3 Weeks Regimen) and Epoch 1 Week 8 (Every 4 Weeks Regimen).

Number of subjects who remained on study to reach full dose. Monthly Dose Equivalent (g/month) is defined as: Full dose in mL \* 1g/10mL / Dose Interval in weeks \* 4.348125 weeks/month and is averaged per subject. Monthly Dose Equivalent (g/kg/month) is defined as: Full dose in mL \* 1g/10mL / Subject's weight in kg at baseline / Dose Interval in weeks \* 4.348125 weeks/month and is averaged per subject.

Duration of infusion(s) per dose will be calculated as the sum of each infusion time for study drug per dose.

Listings of IP exposure and compliance will be provided using the Safety Analysis Set.

## 6.8 Pharmacokinetic, Pharmacodynamic, and Biomarker Analyses

## 6.8.1 Pharmacokinetic Analysis

Analyses for trough serum IgG are described in Section 6.6.3. Additional analysis may be conducted and will be described in a separate pharmacokinetic/pharmacodynamic data analysis plan if applicable.

# 6.8.2 Pharmacodynamic Analysis

Not applicable.

## 6.8.3 **Biomarker Analysis**

Not applicable.

# 6.9 Patient Reported Outcomes (PROs) and Health Care Utilization Endpoints Analysis

## 6.9.1 PRO Analysis

Not applicable.

## 6.9.2 Health Care Utilization Analysis

Not applicable.

## 6.10 Other Analyses

## 1. Time to MMN worsening

Time to MMN worsening is defined as time from the date of the first SC administration of TAK-771 to the date of MMN worsening (where MMN worsening is defined as "Lack of Efficacy" or "Progressive Disease" of primary reason off study treatment). For subjects who worsened in Epoch 1, time to MMN worsening will be calculated as:

Date of treatment end – date of initial dose of IP in Epoch 1 + 1.

Subjects who did not worsening in Epoch 1 will be censored with time to censoring calculated as:

Date of Epoch 1 discontinuation/completion – date of initial dose of IP in Epoch 1 + 1.

In the analysis through Epoch1 and Epoch2, for subjects who worsened, time to worsening will be calculated as:

In the second interim analysis: Date of treatment end of Epoch 2 (The first 6 months of Epoch 2) – date of initial dose of IP in Epoch 1+1.

In the final analysis: Date of treatment end of Epoch 2 (The first 6 months of Epoch 2 or Epoch 2 continued) – date of initial dose of IP in Epoch 1 + 1.

Subjects who did not worsening in Epoch 1 and Epoch 2 will be censored with time to censoring calculated as:

In the second interim analysis: Date of discontinuation/completion of Epoch 2 (The first 6 months of Epoch 2) – date of initial dose of IP in Epoch 1 + 1.

In the final analysis: Last date of discontinuation/completion of Epoch 2 (The first 6 months of Epoch 2 or Epoch 2 continued) – date of initial dose of IP in Epoch 1 + 1.

The statistics presented will include but are not limited to:

- number of subjects included in the analysis
- number of subjects with event
- number of subjects censored
- percentiles (25th, 50th and 75th, if calculable), minimum and maximum for the cumulative incidence (1-survival) function, estimated using the Kaplan-Meier method

Additionally, the cumulative incidence (1-survival) function will be estimated using Kaplan-Meier curves, where the vertical axis will represent the cumulative risk of experiencing a worsening and the number of subjects at-risk over time will be displayed.

#### 6.11 **Interim Analyses**

Two formal interim data analysis to support the Japanese New Drug Application submission will be completed. Both will summarize efficacy and safety of treatment with TAK-771 in Japanese subjects with CIDP/MMN. The first interim analysis will be conducted when the last subject has reached the End of Epoch 1 visit. The second interim analysis will be conducted when the last subject has reached the visit of Week 24 in Epoch 2. The first and the second interim clinical study reports summarizing data will be prepared based on these results of analyses. No adaptive design or data monitoring committee is planned for this study.

In the first interim analysis, the analysis will be performed with data at time points up to the End of Epoch 1. The data listing will include data after the End of Epoch 1.

In the second interim analysis, the analysis will be performed with data at time points up to the Week 24 in Epoch 2. The data listing will include data after the Week 24 in Epoch 2.

In the final analysis, the analysis will be performed with all Epoch 2 data.

# Data Monitoring Committee/Internal Review Committee/ [Other Data Review 6.12 Review, Review **Committees**

No Data Monitoring Committee or Internal Review Committee is planned.

#### 7.0 REFERENCES

- [1] Lewis, R. A., Cornblath, D. R., Hartung, H. P., Sobue, G., Lawo, J. P., Mielke, O., Durn, B. L., Bril, V., Merkies, I. S. J., Bassett, P., Cleasby, A. & Schaik, I. N. 2020. Placebo effect in chronic inflammatory demyelinating polyneuropathy: The PATH study and a systematic review. *Journal of the Peripheral Nervous System*, 25, 230-237.
- [2] Matsui, N. 2012. Multifocal motor neuropathy: current review of epidemiology and treatment. *Rinsho shinkeigaku = Clinical neurology*, 52, 920-2.
- [3] van Nes, S. I., Vanhoutte, E. K., van Doorn, P. A., Hermans, M., Bakkers, M., Kuitwaard, B. Jisab 337-345, in the state of the state K., Faber, C. G. & Merkies, I. S. J. 2011. Rasch-built Overall Disability Scale (R-ODS) for immune-mediated peripheral neuropathies. *Neurology*, 76, 337-345

- properly of Takeda. For non-commercial use only and subject to the applicable of the property of Takeda.

#### 9.0 APPENDIX

## 9.1 Data Handling Conventions

## 9.1.1 General Data Reporting Conventions

TFLs will follow Takeda standards, where applicable, except that footnotes will be printed at the bottom of every output page. IQVIA SOPs and work instructions will apply to all statistical programming, unless otherwise specified in this SAP or the corresponding TFL shells document. Listings will be sorted by cohort, and subject identification number, unless otherwise specified. Both derived and non-derived data, if available, will be displayed in listings.

#### 9.1.2 **Definition of Baseline**

Definition of baseline is described in Section 6.1.

#### 9.1.3 Definition of Visit Windows

For statistical analysis purposes, all efficacy assessments will be assigned to an analysis visit window. Unless otherwise specified for an analysis, the following will apply:

- Assessments will be assigned based on the date the assessment was performed regardless of the completed CRF page.
- Study day will be calculated as: date of assessment date of first dose + 1. The date of the administration 10% IGI will be used as the date of first dose.
- If two or more assessments fall within the same visit window, then the assessment that is closest to the target study day will be used for analysis. If two or more assessments are equidistant from a planned target study day, then the most recent assessment will be used for analysis.
- If there is no assessment within a visit window, then the assessment for that planned study visit will be a considered as missing.

Analysis visit windows are presented for:

- Epoch 1 Efficacy assessments:
  - 2-week regimen (Table 3)
  - o 3-week regimen (Table 4)
  - o 4-week regimen (Table 5)
- Epoch 2 Efficacy assessments:
  - o 2-week regimen (Table 6)
  - o 3-week regimen (Table 7)
  - o 4-week regimen (Table 8)

Table 3 Epoch 1 Analysis Windows for Efficacy Assessments in Subjects with SC Dosing Every 2 Weeks

| Analysis Visit | +/-28) 14 +/-3) 05 +/-3) 89 +/-3) | Epoch 1 Relative Start Day -70 -17 2 109 IRC Sum Scor -17 | Epoch 1 Relative End Day -18 1 108 E1 Last Visit re, GNDS 1 108 | Other Assignment Criteria If E1 relative day is missing and collected visit indicates SCREENING If E1 relative day is missing and collected visit indicates BASELINE If E1 relative day is missing and collected visit indicates E1 and week number ≤ 15 If E1 relative day is missing and collected visit indicates E1 and week number > 15 Last data among E1INT and E0E1 If E1 relative day is missing and collected visit indicates BASELINE If E1 relative day is missing and collected visit indicates BASELINE If E1 relative day is missing and collected visit indicates BASELINE |
|---|---|---|---|---|
| INCAT SCREENING | 42<br>+/-28)<br>14<br>+/-3)<br>05<br>+/-3)<br>89<br>+/-3)<br><b>n, R-ODS, M</b><br>14<br>+/-3)<br>05<br>+/-3) | -17 2 109 IRC Sum Scot | 1 108 E1 Last Visit re, GNDS | If E1 relative day is missing and collected visit indicates SCREENING If E1 relative day is missing and collected visit indicates BASELINE If E1 relative day is missing and collected visit indicates E1 and week number ≤ 15 If E1 relative day is missing and collected visit indicates E1 and week number > 15 Last data among E1INT and EoE1 If E1 relative day is missing and collected visit indicates BASELINE |
| (+/ BASELINE | +/-28) 14 +/-3) 05 +/-3) 89 +/-3) <b>n, R-ODS, M</b> 14 +/-3) 05 +/-3) | -17 2 109 IRC Sum Scot | 1 108 E1 Last Visit re, GNDS | indicates SCREENING If E1 relative day is missing and collected visit indicates BASELINE If E1 relative day is missing and collected visit indicates E1 and week number ≤ 15 If E1 relative day is missing and collected visit indicates E1 and week number > 15 Last data among E1INT and E0E1 If E1 relative day is missing and collected visit indicates BASELINE |
| E1INT 10 (+// E0E1 18 (+// L0E1/6M Hand Grip Strength, BASELINE -1/(+// E1INT 10 (+// E0E1 18 | +/-3) 05 +/-3) 89 +/-3) <b>n, R-ODS, M</b> 14 +/-3) 05 +/-3) | 2<br>109<br>IRC Sum Scot | 108 E1 Last Visit re, GNDS | indicates BASELINE If E1 relative day is missing and collected visit indicates E1 and week number ≤ 15 If E1 relative day is missing and collected visit indicates E1 and week number > 15 Last data among E1INT and EoE1 If E1 relative day is missing and collected visit indicates BASELINE |
| (+/2 EoE1 18 (+/2 EoE1/6M | +/-3) 89 +/-3) 1, R-ODS, M 14 +/-3) 05 +/-3) | 109<br>IRC Sum Scot<br>-17 | E1 Last<br>Visit | indicates E1 and week number ≤ 15 If E1 relative day is missing and collected visit indicates E1 and week number > 15 Last data among E1INT and E0E1 If E1 relative day is missing and collected visit indicates BASELINE |
| EoE1 18 (+/ LoE1/6M Hand Grip Strength, BASELINE -1/ (+/ E1INT 10 (+/ EoE1 18 | 89<br>+/-3)<br><b>n, R-ODS, M</b><br>14<br>+/-3)<br>05<br>+/-3) | IRC Sum Scoi | Visit re, GNDS | indicates E1 and week number > 15 Last data among E1INT and E0E1 If E1 relative day is missing and collected visit indicates BASELINE |
| Hand Grip Strength, BASELINE -14 (+) E1INT 10 (+) E0E1 18 | 14<br>+/-3)<br>05<br>+/-3) | -17 | 1 | If E1 relative day is missing and collected visit indicates BASELINE |
| BASELINE -14 (+) E1INT 10 (+) E0E1 18 | 14<br>+/-3)<br>05<br>+/-3) | -17 | 1 | indicates BASELINE |
| E1INT 10 (+//<br>E0E1 18 | +/-3)<br>05<br>+/-3) | | , , , | indicates BASELINE |
| (+,<br>EoE1 18 | +/-3) | 2 | 108 | If E1 relative day is missing and collected visit |
| | 89 | | | indicates E1 and week number ≤ 15 |
| LoE1/6M | +/-3) | 109 | £1 Last<br>Visit | If E1 relative day is missing and collected visit indicates E1 and week number > 15 |
| | | (0) | | Last data among E1INT and EoE1 |
| LoE1/6M (+) | , non.co | | | |

Table 4 Epoch 1 Analysis Windows for Efficacy Assessments in Subjects with SC Dosing Every 3 Weeks

Table 5 Epoch 1 Analysis Windows for Efficacy Assessments in Subjects with SC Dosing Every 4 Weeks

| 73.76.1 m | Epoch 1<br>Relative<br>Target Day | Epoch 1<br>Relative<br>Start Day | Epoch 1<br>Relative<br>End Day | Other Assignment Criteria |
|---|---|---|---|---|
| INCAT | _ | - | | 2016 |
| SCREENING | -42<br>(+/-28) | -70 | -18 | If E1 relative day is missing and collected vi<br>in SCREENING |
| BASELINE | -14<br>(+/-3) | -17 | 1 | If E1 relative day is missing and collected visindicates BASELINE |
| E1INT | 112<br>(+/-3) | 2 | 115 | If E1 relative day is missing and collected visindicates E1 and week number ≤ 16 |
| EoE1 | 196 (+/-3) | 116 | E1 Last<br>Visit | If E1 relative day is missing and collected vi<br>indicates E1 and week number > 16 |
| LoE1/6M | | | | Last data among E1INT and EoE1 |
| | ength, R-ODS, M | RC Sum Scor | re, GNDS | 250 |
| BASELINE | -14<br>(+/-3) | -17 | 1 | If E1 relative day is missing and collected vi<br>indicates BASELINE |
| E1INT | 112<br>(+/-3) | 2 | 115 | If E1 relative day is missing and collected vi<br>indicates E1 and week number ≤ 16 |
| EoE1 | 196 | 116 | E1 Last<br>Visit | If E1 relative day is missing and collected vi<br>indicates E1 and week number > 16 |
| LoE1/6M | | (0) | | Last data among E1INT and EoE1 |
| | (+/-3) | | | |

Table 6 Epoch 2 Analysis Windows for Efficacy Assessments (Dosing Every 2 Weeks)

| | Epoch 2<br>Relative <sup>a</sup> | Epoch 2<br>Relative | Epoch 2<br>Relative | |
|---|---|---|---|---|
| Analysis Visit | Target Day | Start Day | End Day | Other Assignment Criteria |
| INCAT, Hand gr | ip strength (Fo | r MMN subje | cts) | |
| E2W4 | 29(+/-3) | 26 | 43 | If E2 relative day is missing and collected visit indicates E2 and week number 4 |
| E2W8 | 57(+/-3) | 44 | 71 | If E2 relative day is missing and collected visit indicates E2 and week number 8 |
| E2W12 | 85(+/-3) | 72 | 99 | If E2 relative day is missing and collected visit indicates E2 and week number 12 |
| E2W16 | 113(+/-3) | 100 | 127 | If E2 relative day is missing and collected visit indicates E2 and week number 16 |
| E2W20 | 141(+/-3) | 128 | 155 | If E2 relative day is missing and collected visit indicates E2 and week number 20 |
| E2W24/Eo6M | 169(+/-3) | 156 | 183 | If E2 relative day is missing and collected visit indicates Eo6M or (E2 and week number 24) |
| LoE2/6M | | | 388 | Last data among E2W4, E28W, E2W12,<br>E2W16, E2W20 and E2W24/E06M |
| E2C3M | 85(+/-3) | 1 | 88 | |
| E2C6M | 169(+/-3) | 89 | 172 | |
| E2C9M | 253(+/-3) | 173 | 256 | |
| E2C12M | 337(+/-3) | 257 | 340 | |
| E2C15M | 421(+/-3) | 341 | 424 | |
| E2C18M | 505(+/-3) | 425 | 508 | |
| E2C21M | 589(+/-3) | 509 | 592 | |
| E2C24M | 673(+/-3) | 593 | 676 | |
| E2C27M | 357(+/-3) | 677 | 760 | |
| LoE2C | | | | Last data among E2CnM (n: 3, 6, 9,) |
| EoS | | | | Last data throughout the study (Epoch 1 to Epoch 2) |
| Hand grip streng | th (For CIDP s | ubjects), R-O | DS, MRC sum | score, GNDS |
| E2W12 | 85(+/-3) | 72 | 99 | If E2 relative day is missing and collected visit indicates E2 and week number 12 |
| E2W24/Eo6M | 169(+/-3) | 156 | 183 | If E2 relative day is missing and collected visit indicates Eo6M or (E2 and week number 24) |
| LoE2/6M | | | | Last data among E2W12 and E2W24/Eo6M |
| E2C3M | 85(+/-3) | 1 | 88 | |
| E2C6M | 169(+/-3) | 89 | 172 | |

**Epoch 2 Analysis Windows for Efficacy Assessments (Dosing Every** Table 6 2 Weeks)

| | Epoch 2 | Epoch 2 | Epoch 2 | |
|---|---|---|---|---|
| Analysis Visit | Relative <sup>a</sup><br>Target Day | Relative<br>Start Day | Relative<br>End Day | Other Assignment Criteria |
| E2C9M | 253(+/-3) | 173 | 256 | 201 |
| E2C12M | 337(+/-3) | 257 | 340 | 1,00 |
| E2C15M | 421(+/-3) | 341 | 424 | 20/1 |
| E2C18M | 505(+/-3) | 425 | 508 | 2/ |
| E2C21M | 589(+/-3) | 509 | 592 | /\© |
| E2C24M | 673(+/-3) | 593 | 676 | 1.0 |
| E2C27M | 757(+/-3) | 677 | 760 | A. W. |
| LoE2C | 1 | | | Last data among E2CnM (n: 3, 6, 9,) |
| EoS | | | | T + 1 × 0 + 1 /T + 1 1 / |
| of the first infusion | - | | | Last data throughout the study (Epoch 1 to Epoch 2) ed on the date of the first Epoch 2 infusion; the day 2 after 6 months is based on the date of the first infusion is E2 (continued) Day 1. |
| of the first infusion<br>Epoch 2 infusion o | n is E2 Day 1. Ep | | | Epoch 2) ed on the date of the first Epoch 2 infusion; the day |
| of the first infusion | n is E2 Day 1. Ep | ooch 2 relative | | Epoch 2) ed on the date of the first Epoch 2 infusion; the day |

<sup>&</sup>lt;sup>a</sup> Epoch 2 relative day for Epoch 2 until the first 6 months is based on the date of the first Epoch 2 infusion; the day of the first infusion is E2 Day 1. Epoch 2 relative day for Epoch 2 after 6 months is based on the date of the first

Table 7 Epoch 2 Analysis Windows for Efficacy Assessments (Dosing Every 3 Weeks)

| | | E 10 | E 1.0 | |
|---|---|---|---|---|
| | Epoch 2<br>Relative <sup>a</sup> | Epoch 2<br>Relative | Epoch 2<br>Relative | 405 |
| Analysis Visit | Target Day | Start Day | End Day | Other Assignment Criteria |
| INCAT, Hand gr | rip strength (Fo | r MMN subje | cts) | 90, |
| E2W3 | 22(+/-3) | 17 | 43 | If E2 relative day is missing and collected visit indicates E2 and week number 3 |
| E2W9 | 64(+/-3) | 44 | 74 | If E2 relative day is missing and collected visit indicates E2 and week number 9 |
| E2W12 | 85(+/-3) | 75 | 95 | If E2 relative day is missing and collected visit indicates E2 and week number 12 |
| E2W15 | 106(+/-3) | 96 | 127 | If E2 relative day is missing and collected visit indicates E2 and week number 15 |
| E2W21 | 148(+/-3) | 128 | 158 | If E2 relative day is missing and collected visit indicates E2 and week number 21 |
| E2W24/Eo6M | 169(+/-3) | 159 | 179 | HE2 relative day is missing and collected visit<br>indicates Eo6M or (E2 and week number 24) |
| LoE2/6M | | | OULA | Last data among E2W4, E28W, E2W12,<br>E2W16, E2W20 and E2W24/E06M |
| E2C3M | 85(+/-5) | 1 | 900 | |
| E2C6M | 169(+/-5) | 91 | 174 | |
| E2C9M | 253(+/-5) | 175 | 258 | |
| E2C12M | 337(+/-5) | 259 | 342 | |
| E2C15M | 421(+/-5) | 343 | 426 | |
| E2C18M | 505(+/-5) | 427 | 510 | |
| E2C21M | 589(+/-5) | 511 | 594 | |
| E2C24M | 673(+/3) | 595 | 678 | |
| E2C27M | 757(+7-5) | 679 | 762 | |
| LoE2C | .0 | | | Last data among E2CnM (n: 3, 6, 9,) |
| EoS | • | | | Last data throughout the study (Epoch 1 to Epoch 2) |

**Epoch 2 Analysis Windows for Efficacy Assessments (Dosing Every** Table 7 3 Weeks)

| Analysis Visit | Epoch 2<br>Relative <sup>a</sup><br>Target Day | Epoch 2<br>Relative<br>Start Day | Epoch 2<br>Relative<br>End Day | Other Assignment Criteria |
|---|---|---|---|---|
| Hand grip stren | - | • | • | |
| E2W12 | 85(+/-5) | 75 | 95 | If E2 relative day is missing and collected visit indicates E2 and week number 12 |
| E2W24/Eo6M | 169(+/-5) | 159 | 179 | If E2 relative day is missing and collected visit indicates Eo6M or (E2 and week number 24) |
| LoE2/6M | | | | Last data among E2W12 and E2W24/Eo6M |
| E2C3M | 85(+/-5) | 1 | 90 | 1,40 |
| E2C6M | 169(+/-5) | 91 | 174 | C. |
| E2C9M | 253(+/-5) | 175 | 258 | NIO. |
| E2C12M | 337(+/-5) | 259 | 342 | a) |
| E2C15M | 421(+/-5) | 343 | 426 | -0 |
| E2C18M | 505(+/-5) | 427 | 510 | <u></u> |
| E2C21M | 589(+/-5) | 511 | 594 | |
| E2C24M | 673(+/-5) | 595 | 678 | |
| E2C27M | 757(+/-5) | 679 | 762) | |
| LoE2C | | | 72 | Last data among E2CnM (n: 3, 6, 9,) |
| EoS | | (i) | | Last data throughout the study (Epoch 1 to Epoch 2) |
| of the first infusion | .* | | day for Epoch | d on the date of the first Epoch 2 infusion; the d<br>2 after 6 months is based on the date of the first<br>infusion is E2 (continued) Day 1. |

<sup>&</sup>lt;sup>a</sup> Epoch 2 relative day for Epoch 2 until the first 6 months is based on the date of the first Epoch 2 infusion; the day of the first infusion is E2 Day 1. Epoch 2 relative day for Epoch 2 after 6 months is based on the date of the first

Table 8 Epoch 2 Analysis Windows for Efficacy Assessments (Dosing Every 4 Weeks)

| | Epoch 2<br>Relative <sup>a</sup> | Epoch 2<br>Relative | Epoch 2<br>Relative | ZO! |
|---|---|---|---|---|
| Analysis Visit | Target Day | Start Day | End Day | Other Assignment Criteria |
| INCAT, Hand gr | rip strength (Fo | r MMN subje | cts) | 90, |
| E2W4 | 29(+/-3) | 26 | 43 | If E2 relative day is missing and collected visit indicates E2 and week number 4 |
| E2W8 | 57(+/-3) | 44 | 71 | If E2 relative day is missing and collected visit indicates E2 and week number 8 |
| E2W12 | 85(+/-3) | 72 | 99 | If E2 relative day is missing and collected visit indicates E2 and week number 12 |
| E2W16 | 113(+/-3) | 100 | 127 | If E2 relative day is missing and collected visit indicates E2 and week number 16 |
| E2W20 | 141(+/-3) | 128 | 155 | If E2 relative day is missing and collected visit indicates E2 and week number 20 |
| E2W24/Eo6M | 169(+/-3) | 156 | 183 | HE2 relative day is missing and collected visit<br>indicates Eo6M or (E2 and week number 24) |
| LoE2/6M | | | OULA | Last data among E2W4, E28W, E2W12, E2W16, E2W20 and E2W24/E06M |
| E2C3M | 85(+/-7) | 1 | 92 | |
| E2C6M | 169(+/-7) | 93 | 176 | |
| E2C9M | 253(+/-7) | 177 | 260 | |
| E2C12M | 337(+/-7) | 261 | 344 | |
| E2C15M | 421(+/-7) | 345 | 428 | |
| E2C18M | 505(+/-7) | 429 | 512 | |
| E2C21M | 589(+/-7) | 513 | 596 | |
| E2C24M | 673(+/-7) | 597 | 680 | |
| E2C27M | 757(+/-7) | 681 | 764 | |
| LoE2C | 0 | | | Last data among E2CnM (n: 3, 6, 9,) |
| EoS | | | | Last data throughout the study (Epoch 1 to Epoch 2) |

**Epoch 2 Analysis Windows for Efficacy Assessments (Dosing Every** Table 8 4 Weeks)

| Analysis Visit | Epoch 2<br>Relative <sup>a</sup><br>Target Day | Epoch 2<br>Relative<br>Start Day | Epoch 2<br>Relative<br>End Day | Other Assignment Criteria |
|---|---|---|---|---|
| Hand grip stren | | • | | |
| E2W12 | 85(+/-3) | 72 | 99 | If E2 relative day is missing and collected vis indicates E2 and week number 12 |
| E2W24/Eo6M | 169(+/-3) | 156 | 183 | If E2 relative day is missing and collected vis indicates Eo6M or (E2 and week number 24) |
| LoE2/6M | | | | Last data among E2W12 and E2W24/E06M |
| E2C3M | 85(+/-7) | 1 | 92 | 1,10 |
| E2C6M | 169(+/-7) | 93 | 176 | 20 |
| E2C9M | 253(+/-7) | 177 | 260 | 100 |
| E2C12M | 337(+/-7) | 261 | 344 | 6), |
| E2C15M | 421(+/-7) | 345 | 428 | -9 |
| E2C18M | 505(+/-7) | 429 | 512 | |
| E2C21M | 589(+/-7) | 513 | 596 | |
| E2C24M | 673(+/-7) | 597 | 680 | |
| E2C27M | 757(+/-7) | 681 | 7.64) | |
| LoE2C | | | 100 | Last data among E2CnM (n: 3, 6, 9,) |
| EoS | | ,cia | | Last data throughout the study (Epoch 1 to Epoch 2) |
| | n is E2 Day 1. E | | day for Epoch | ed on the date of the first Epoch 2 infusion; the 2 after 6 months is based on the date of the first infusion is E2 (continued) Day 1. |

<sup>&</sup>lt;sup>a</sup> Epoch 2 relative day for Epoch 2 until the first 6 months is based on the date of the first Epoch 2 infusion; the day of the first infusion is E2 Day 1. Epoch 2 relative day for Epoch 2 after 6 months is based on the date of the first

## 9.1.4 Repeated or Unscheduled Assessments of Safety Parameters

If a subject has repeated assessments before initial dose of IP, then the most recent assessment value will be used as baseline in analysis/summaries involving baseline.

If a subject has repeated assessments after initial dose of IP (repeated post-baseline assessments), then the most recent assessment value will be used in analysis/summaries involving post-baseline.

Unscheduled assessments (i.e., assessments not done at a planned visit) will used only in summaries of abnormalities or toxicities (not otherwise).

All assessments, including repeated and unscheduled assessments, will be presented in the subject data listings.

## 9.1.5 Handling of Missing, Unused, and Spurious Data

This section provides a general plan for handling of missing data, unused and spurious data. Specifics regarding handling are addressed in specific endpoint analysis sections.

Data that appear to be spurious (e.g., outliers, incompatible with life) will be queried by Clinical Data Management and then either corrected or explained in the CSR if not correctable. Outliers will not be excluded from analysis unless otherwise specified. Any exclusion of data from analysis will be appropriately footnoted in the relevant TFLs.

# 9.1.6 Missing Date of Investigational Product

If the date of the last dose of IP is missing for a subject in the Safety analysis set, then all efforts will be made by the study sponsor, or on behalf of the sponsor, to obtain the date from the study investigator. If the date cannot be obtained despite all efforts, then the last visit date when IP was dispensed will be used in the calculation of treatment duration.

That is, if last dose date is missing, then last visit in Treatment Period date will be used.

# 9.1.7 Missing Date Information for Prior or Concomitant Medications (Therapies/Procedures)

For prior or concomitant medications (and/or therapies/procedures), incomplete (fully or partially missing) start date and/or stop date of mediation will be imputed. When the start date and the stop date are both incomplete for a subject, impute the start date first using the imputation approach described in the subsequent sections.

## 91.7.1 Incomplete Start Date

The following rules will be applied to impute the missing numerical fields. If the stop date is complete and the imputed start date is after the stop date, then the start date will be imputed using the stop date.

## 9.1.7.1.1 Missing Day and Month

- If the year of the incomplete start date is the same as the year of the date of the first dose of IP, then the day and month of the date of the first dose of IP will be assigned to the missing fields
- If the year of the incomplete start date is before the year of the date of the first dose of IP, then December 31 will be assigned to the missing fields
- If the year of the incomplete start date is after the year of the date of the first dose of IP, then 01 January will be assigned to the missing fields

## 9.1.7.1.2 Missing Month Only

• The day will be treated as missing and both month and day will be replaced according to the above procedure

## 9.1.7.1.3 Missing Day Only

- If the month and year of the incomplete start date are the same as the month and year of the date of the first dose of IP, then the day of the date of the first dose of IP will be assigned to the missing day
- If either the year is before the year of the date of the first dose of IP, or if both years are the same but the month is before the month of the date of the first dose of IP, then the last day of the month will be assigned to the missing day
- If either the year is after the year of the date of the first dose of IP, or if both years are the same but the month is after the month of the date of the first dose of IP, then the first day of the month will be assigned to the missing day

# 9.1.7.2 Incomplete Stop Date

The following rules will be applied to impute the missing numerical fields. If the date of the last dose of IP is missing, then replace it with the last visit date. If the imputed stop date is before the (imputed or non-imputed) start date, then the imputed stop date will be equal to the start date.

If imputation of an incomplete stop date is required for calculating duration, and both the start date and the stop date are incomplete for a subject, then the start date will be imputed first.

A completely missing stop date will be interpreted as ongoing.

# 9.1.7.2.1 Missing Day and Month

- If the year of the incomplete stop date is the same as the year as of the date of the last dose of IP, then the day and month of the date of the last dose of IP will be assigned to the missing fields
- If the year of the incomplete stop date is before the year of the date of the last dose of IP, then 31 December will be assigned to the missing fields

• If the year of the incomplete stop date is after the year of the date of the last dose of IP, then 01 January will be assigned to the missing fields

## 9.1.7.2.2 Missing Month Only

• The day will be treated as missing and both month and day will be replaced according to the above procedure

## 9.1.7.2.3 Missing Day Only

- If the month and year of the incomplete stop date are the same as the month and year of the date of the last dose of IP, then the day of the date of the last dose of IP will be assigned to the missing day
- If the year is before the year of the date of the last dose of IP, or if both years are the same but the month is before the month of the date of the last dose of IP, then the last day of the month will be assigned to the missing day
- If the year is after the year of the last dose of IP, or if both years are the same but the month is after the month of the date of the last dose of IP, then the first day of the month will be assigned to the missing day

## 9.1.8 Missing Date Information for Adverse Events

The following approaches will be applied:

- To facilitate categorization of AEs as treatment emergent, imputation of dates can be used
- If an AE start date is completely missing, then the AE will be considered treatment-emergent in Epoch 1
- For AEs with partial start dates, non-missing date parts will be used to determine if the AE is treatment-emergent or not. If a determination cannot be made using the non-missing date parts as to when the AE occurred relative to IP (eg, AE start year and month are the same as the year and month of the first dose of IP), then the AE will be classified as treatment-emergent
- For AEs, the default is to only impute incomplete (i.e., partially missing) start dates. Incomplete stop dates may also be imputed when calculation of the duration of an AE is required per the protocol
- If imputation of an incomplete stop date is required, and both the start date and the stop date are incomplete for a subject, impute the start date first

## 9.1.8.1 Incomplete Start Date

Rules in Section 9.1.7.1 apply.

## 9.1.8.2 Incomplete Stop Date

Rules in Section 9.1.7.2 apply.

## 9.1.9 Missing Date Information for First Symptoms

Incomplete (fully or partially missing) date of first symptoms will be imputed. Rules in Section 9.1.7.1 apply.

## 9.1.10 Missing Date Information for Diagnosis

Incomplete (fully or partially missing) date of diagnosis will be imputed. Rules in Section 9.1.7.1 apply.

## 9.1.11 Missing Severity Assessment for Adverse Events

If severity is missing for an AE starting prior to the date of the first dose of IP, then a severity of "Mild" will be assigned. If the severity is missing for an AE starting on or after the date of the first dose of IP, then a severity of "Severe" will be assigned.

If a subject experiences more than one AE categorized under the same preferred term, where one of them is categorized as "severe" and one of them is categorized as "unknown", then the severity of this AE will be counted as "severe".

If a subject experiences more than one AE categorized under the same preferred term, where one of them is categorized as "mild" or "moderate" and one of them is categorized as "unknown", then the severity of this AE will be counted as "unknown".

The imputed values for severity assessment will be used for summaries, while both the actual and the imputed values will be used in subject data listings.

## 9.1.12 Missing Seriousness of Adverse Events

AEs of unknown seriousness will be tabulated as SAEs in summaries; however, every effort will be made to avoid study data lock with AEs for which a determination of seriousness is missing.

# 9.1.13 Missing Relationship to Investigational Product for Adverse Events

If the relationship to IP is missing for an AE starting on or after the date of the first dose of IP, then a causality of "related" will be assigned. The imputed values for relationship to IP will be used for incidence summaries, while both the actual and the imputed values will be presented in data listings.

#### 9.1.14 **Character Values of Clinical Laboratory Variables**

in sofuse Laboratory measurements will be presented in SI units, unless otherwise specified for an analysis. If a laboratory result is expected to have a numeric value, but the data which are received include a special character such as ">" or "<", then the result will be assumed to lie outside the range of quantitation (example: if the data is < 30 or <= 30, the result will assume to be 29).

Tables based on a dichotomous or categorical grouping, including but not limited to shift tables, Acr., naries is esigned to esigned to the end of the en will place such data appropriately prior to removal of the special character, so that particularly low or high values remain recognized as such. For quantitative summaries by time-point or visit, the numeric part of such a result will be used, unless the table is designed to include explicit

## 9.2 Definition of AESIs

Definition information for AESIs in MedDRA ver.26.0 is provided in the following tables. Since there is no change in the definition of AESIs in table 9 between MedDRA ver. 26.0 and ver. 27.0, the same definitions will also be used in MedDRA ver. 27.0.

Table 9 Adverse Events of Special Interest

| Display Category | Display Term | AEDECOD in Upper<br>Case | PT Code<br>(MedDRA<br>ver.26.0) | Additional<br>Conditions |
|---|---|---|---|---|
| Allergic Reactions | Urticaria | URTICARIA | 10046735 | |
| | New-onset<br>bronchospasm | BRONCHOSPASM | 10006482 | |
| | Oedema of tongue, lips, face (angioedema) | Refer to Table 9.1 : Oed lips, face (angioedema) | | |
| | Anaphylaxis | Refer to Table 9.2 : An | | |
| | Stevens-Johnson<br>syndrome | STEVENS-<br>JOHNSON<br>SYNDROME | 10042033 | |
| | Erythema multiforme | ERYTHEMA<br>MULTIFORME | 10015218 | |
| | Toxic epidermal necrolysis | FOXIC 10044223<br>EPIDERMAL<br>NECROLYSIS | | |
| Immune complex mediated reactions - | Persistent induration or nodule | Refer to Table 9.3 : Persistent induration or nodule | | Duration > 48<br>hours (> 2 days) |
| Local | Excessive inflammation | Refer to Table 9.4 : Exc<br>inflammation | Severity = "SEVERE" | |
| | Tissue necrosis/ulceration at the site of administration | Refer to Table 9.5 : Tis necrosis/ulceration | | |
| Aega. For | Dystrophic or fibrotic changes at the site of administration | Refer to Table 9.6 : Dystrophic or fibrotic changes | | |
| 1 2 4 6 9 s. | Pigmented skin changes<br>at the site of drug<br>administration | Refer to Table 9.7 :Pigmented skin changes | | |
| Immune complex | Arthritis | ARTHRITIS | 10003246 | |
| mediated reactions - | Vasculitis (purpuric | VASCULITIS | 10047115 | |
| Systemic | rash) | Refer to Table 9.8 : Ras | sh | |
| | | Refer to Table 9.9 : Pur | pura | |
| | Glomerulonephritis | HAEMATURIA | 10018867 | |
| | | Refer to Table 9.10 : No | ephritis | |

#### **Adverse Events of Special Interest** Table 9

| Display Category | Display Term | AEDECOD in Upper<br>Case | PT Code<br>(MedDRA<br>ver.26.0) | Additional<br>Conditions |
|---|---|---|---|---|
| Thrombotic/embolic | Arterial | Refer to Table 9.11 : A | rterial | 01 |
| events | Venous | Refer to Table 9.12 : V | Refer to Table 9.12 : Venous | |
| | Vessel<br>unspecified/unknown | Refer to Table 9.13 : Vessel<br>unspecified/unknown | | olico |
| Table 9.1 Oed | lema of tongue, lips, fa | ice (angioedema) | ine | ,0, |
| AFDECOD | | | PT Code | |

#### Oedema of tongue, lips, face (angioedema) Table 9.1

| AEDECOD | | PT Code |
|---------------|------|----------|
| Angioedema | ·(©) | 10002424 |
| Face oedema | 10, | 10016029 |
| Lip oedema | 350 | 10024558 |
| Tongue oedema | -10 | 10043967 |

#### Anaphylaxis Table 9.2

| AEDECOD | 119 | PT Code |
|-----------------------|------|----------|
| Anaphylactic reaction | . 7 | 10002198 |
| Anaphylactic shock | , C) | 10002199 |

#### Persistent induration or nodule Table 9.3

| AEDECOD | PT Code |
|--------------------------------|----------|
| Injection site induration | 10022075 |
| Infusion site induration | 10053482 |
| Administration site induration | 10075939 |
| Injection site nodule | 10057880 |
| Infusion site nodule | 10065484 |
| Administration site nodule | 10075765 |

**Table 9.4** Excessive inflammation

| AEDECOD | PT Code |
|----------------------------------------|----------|
| Injection site inflammation | 10022078 |
| Infusion site inflammation | 10056270 |
| Injection site joint inflammation | 10064111 |
| Administration site inflammation | 10074704 |
| Administration site joint inflammation | 10075946 |
| Infusion site joint inflammation | 10076074 |
| Injection site joint swelling | 10049260 |
| Injection site swelling | 10053425 |
| Infusion site swelling | 10053505 |
| Administration site swelling | 10075107 |
| Infusion site joint swelling | 10076078 |
| Injection site pain | 10022086 |
| Injection site joint pain | 10049261 |
| Infusion site pain | 10053483 |
| Administration site pain | 10058049 |
| Administration site joint pain | 10075948 |

Table 9.5 Tissue necrosis/ulceration

| AEDECOD | PT Code |
|------------------------------|----------|
| Injection site necrosis | 10022082 |
| Infusion site necrosis | 10065478 |
| Administration site necrosis | 10075956 |
| Injection site ulcer | 10022105 |
| Infusion site ulcer | 10054995 |
| Administration site ulcer | 10075108 |

## Table 9.6 Dystrophic or fibrotic changes

| AEDECOD | PT Code |
|----------------------------------|----------|
| Injection site fibrosis | 10022064 |
| Infusion site fibrosis | 10065462 |
| Administration site fibrosis | 10075934 |
| Injection site dysaesthesia | 10069124 |
| Administration site dysaesthesia | 10075930 |
| Infusion site dysaesthesia | 10076067 |

## Table 9.7 Pigmented skin changes

| AEDECOD | PT Code |
|------------------------------------|----------|
| Injection site discolouration | 19051572 |
| Infusion site discolouration | 10065460 |
| Administration site discolouration | 10075098 |

## Table 9.8 Rash

| AEDECOD | PT Code |
|-----------------------------------|----------|
| Rash | 10037844 |
| Rash erythematous | 10037855 |
| Rash follicular | 10037857 |
| Rash macular | 10037867 |
| Rash maculo-papular | 10037868 |
| Rash morbilliform | 10037870 |
| Rash neonatal | 10037871 |
| Rash papular | 10037876 |
| Rash papulosquamous | 10037879 |
| Rash pruritic | 10037884 |
| Rash scarlatiniform | 10037890 |
| Rash vesicular | 10037898 |
| Systemic lupus erythematosus rash | 10042946 |
| Vasculitic rash | 10047111 |
| Rash maculovesicular | 10050004 |
| Mucocutaneous rash | 10056671 |
| Rash rubelliform | 10057984 |
| Exfoliative rash | 10064579 |
| Butterfly rash | 10067982 |
| Paraneoplastic rash | 10074687 |
| Nodular rash | 10075807 |
| Heliotrope rash | 10081454 |

## Table 9.9 Purpura

| AEDECOD | PT Code |
|------------------------------------------------|----------|
| Henoch-Schonlein purpura | 10019617 |
| Purpura | 10037549 |
| Purpura fulminans | 10037556 |
| Purpura neonatal | 10037557 |
| Purpura senile | 10037560 |
| Vascular purpura | 10047097 |
| Palpable purpura | 10056872 |
| Chronic pigmented purpura | 10072726 |
| Hypergammaglobulinaemic purpura of Waldenstrom | 10086403 |

# Table 9.10 Nephritis

| AEDECOD Glomerulonephritis Glomerulonephritis rapidly progressive Lupus nephritis Lupus nephri | Tuble 5126 Trepartors | |
|---|---|---|
| Glomerulonephritis rapidly progressive 10018378 Lupus nephritis 10025140 Fibrillary glomerulonephritis 10068279 Tubulointerstitial nephritis and uveitis syndrome 10069034 Henoch-Schonlein purpura nephritis 10069440 Chronic autoimmune glomerulonephritis 10073016 | AEDECOD | PT Code |
| Lupus nephritis 10025140 Fibrillary glomerulonephritis 10068279 Tubulointerstitial nephritis and uveitis syndrome 10069034 Henoch-Schonlein purpura nephritis 10069440 Chronic autoimmune glomerulonephritis 10073016 | Glomerulonephritis | 10018364 |
| Fibrillary glomerulonephritis 10068279 Tubulointerstitial nephritis and uveitis syndrome 10069034 Henoch-Schonlein purpura nephritis 10069440 Chronic autoimmune glomerulonephritis 10073016 | Glomerulonephritis rapidly progressive | 10018378 |
| Tubulointerstitial nephritis and uveitis syndrome 10069034 Henoch-Schonlein purpura nephritis 10069440 Chronic autoimmune glomerulonephritis 10073016 | Lupus nephritis | 10025140 |
| Henoch-Schonlein purpura nephritis 10069440 Chronic autoimmune glomerulonephritis 10073016 | | 10068279 |
| Chronic autoimmune glomerulonephritis | Tubulointerstitial nephritis and uveitis syndrome | 10069034 |
| | Henoch-Schonlein purpura nephritis | 10069440 |
| Autoimmune nephritis 10077087 Immune-mediated nephritis 10083070 | Chronic autoimmune glomerulonephritis | 10073016 |
| Immune-mediated nephritis 10083070 | Autoimmune nephritis | 10077087 |
| of Takedai. For nonr.co | Immune-mediated nephritis | 10083070 |
| | of Lakedai. | |

Table 9.11 Arterial

| Table 9.11 Arterial | |
|------------------------------------------|----------|
| AEDECOD in Upper Case | PT Code |
| CAROTID ENDARTERECTOMY | 10007692 |
| RETINAL ARTERY EMBOLISM | 10038826 |
| ARTERECTOMY WITH GRAFT REPLACEMENT | 10003140 |
| HYPOTHENAR HAMMER SYNDROME | 10063518 |
| CEREBRAL ARTERY THROMBOSIS | 10008092 |
| PERIPHERAL ARTERIAL OCCLUSIVE DISEASE | 10062585 |
| MESENTERIC ARTERY THROMBOSIS | 10027397 |
| COELIAC ARTERY OCCLUSION | 10069696 |
| ARTERIAL GRAFT | 10061655 |
| CAPSULAR WARNING SYNDROME | 10067744 |
| PERIPHERAL ARTERIAL REOCCLUSION | 10069379 |
| MESENTERIC ARTERY EMBOLISM | 10027395 |
| AORTIC BYPASS | 10057617 |
| ENDARTERECTOMY | 10014648 |
| ACUTE AORTIC SYNDROME | 10074337 |
| CEREBRAL HYPOPERFUSION | 10065384 |
| TRUNCUS COELIACUS THROMBOSIS | 10062363 |
| FEMORAL ARTERY EMBOLISM | 10068365 |
| PERIPHERAL ARTERY THROMBOSIS | 10072564 |
| SUPERIOR MESENTERIC ARTERY SYNDROME | 10054156 |
| STROKE IN EVOLUTION | 10059613 |
| CORONARY ARTERY EMBOLISM | 10011084 |
| ATHERECTOMY | 10063025 |
| ILIAC ARTERY OCCLUSION | 10064601 |
| ATRIAL APPENDAGE CLOSURE | 10079735 |
| CAROTID ARTERY OCCLUSION | 10048964 |
| ARTERIAL OCCLUSIVE DISEASE | 10062599 |
| MESENTERIC ARTERY STENT INSERTION | 10071261 |
| INTRAOPERATIVE CEREBRAL ARTERY OCCLUSION | 10056382 |
| ARTERIOGRAM ABNORMAL | 10061659 |
| CEREBRAL ARTERY EMBOLISM | 10008088 |
| HEPATIC ARTERY EMBOLISM | 10019635 |
| AMAUROSIS | 10001902 |
| ARTERIOGRAM CAROTID ABNORMAL | 10003195 |
| SPINAL ARTERY EMBOLISM | 10049440 |
| SUBCLAVIAN ARTERY OCCLUSION | 10069695 |
| THROMBOEMBOLECTOMY | 10064958 |

Table 9.11 Arterial

| Table 9.11 Afterial | |
|------------------------------------|----------|
| AEDECOD in Upper Case | PT Code |
| CAROTID ARTERY STENT INSERTION | 10066102 |
| PERIPHERAL ENDARTERECTOMY | 10072560 |
| SPLENIC EMBOLISM | 10068677 |
| SPINAL ARTERY THROMBOSIS | 10071316 |
| AORTIC EMBOLUS | 10002897 |
| PERIPHERAL ARTERY BYPASS | 10072561 |
| PERIPHERAL ARTERY STENT INSERTION | 10072562 |
| RETINAL ARTERY THROMBOSIS | 10038831 |
| CAROTID ARTERY THROMBOSIS | 10007688 |
| ANGIOPLASTY | 10002475 |
| BASAL GANGLIA INFARCTION | 10069020 |
| CORONARY ARTERIAL STENT INSERTION | 10052086 |
| HEPATIC ARTERY THROMBOSIS | 10019636 |
| CEREBELLAR ARTERY OCCLUSION | 10053633 |
| THROMBOTIC MICROANGIOPATHY | 10043645 |
| MESENTERIC ARTERIOSCLEROSIS | 10065560 |
| AORTIC THROMBOSIS | 10002910 |
| CAROTID ARTERIAL EMBOLUS | 10007684 |
| MYOCARDIAL INFARCTION | 10028596 |
| ARTERIAL THROMBOSIS | 10003178 |
| TRANSIENT ISCHAEMIC ATTACK | 10044390 |
| PULMONARY ENDARTERECTOMY | 10072893 |
| MYOCARDIAL NECROSIS | 10028602 |
| POSTINFARCTION ANGINA | 10058144 |
| STRESS CARDIOMYOPATHY | 10066286 |
| CEREBROVASCULAR STENOSIS | 10061751 |
| INTRA-AORTIC BALLOON PLACEMENT | 10052989 |
| CAROTID ARTERY BYPASS | 10053003 |
| HEPATIC ARTERY OCCLUSION | 10051991 |
| SPLENIC ARTERY THROMBOSIS | 10074600 |
| AMAUROSIS FUGAX | 10001903 |
| SILENT MYOCARDIAL INFARCTION | 10049768 |
| PERCUTANEOUS CORONARY INTERVENTION | 10065608 |
| CEREBELLAR ARTERY THROMBOSIS | 10008023 |
| VERTEBRAL ARTERY OCCLUSION | 10048965 |
| ARTERECTOMY | 10071026 |
| ACUTE MYOCARDIAL INFARCTION | 10000891 |
| | • |

Table 9.11 Arterial

| AEDECOD in Upper Case | PT Code |
|---------------------------------------------------------|----------|
| BRACHIOCEPHALIC ARTERY OCCLUSION | 10069694 |
| CORONARY ARTERY BYPASS | 10011077 |
| PENILE ARTERY OCCLUSION | 10068035 |
| CEREBROVASCULAR INSUFFICIENCY | 10058842 |
| BLINDNESS TRANSIENT | 10005184 |
| VERTEBRAL ARTERY THROMBOSIS | 10057777 |
| POPLITEAL ARTERY ENTRAPMENT SYNDROME | 10071642 |
| CORONARY ENDARTERECTOMY | 10011101 |
| CORONARY VASCULAR GRAFT OCCLUSION | 10075162 |
| AORTIC SURGERY | 10061651 |
| CORONARY ARTERY REOCCLUSION | 10053261 |
| SUBCLAVIAN ARTERY THROMBOSIS | 10042334 |
| BASILAR ARTERY THROMBOSIS | 10063093 |
| PULMONARY ARTERY THROMBOSIS | 10037340 |
| CORONARY REVASCULARISATION | 10049887 |
| LACUNAR INFARCTION | 10051078 |
| PRECEREBRAL ARTERY THROMBOSIS | 10074717 |
| CORONARY ARTERY OCCLUSION | 10011086 |
| AORTOGRAM ABNORMAL | 10057794 |
| RENAL ARTERY OCCLUSION | 10048988 |
| ISCHAEMIC CEREBRAL INFARCTION | 10060840 |
| PULMONARY ARTERY THERAPEUTIC PROCEDURE | 10063731 |
| MESENTERIC ARTERIAL OCCUUSION | 10027394 |
| RENAL ARTERY ANGIOPLASTY | 10057493 |
| CORONARY ARTERY THROMBOSIS | 10011091 |
| ILIAC ARTERY EMBOLISM | 10021338 |
| CORONARY ANGIOPLASTY | 10050329 |
| CAROTID ANGIOPLASTY | 10071260 |
| CEREBRAL ARTERY OCCLUSION | 10008089 |
| ATHEROSCLEROTIC PLAQUE RUPTURE | 10076604 |
| ARTERIAL STENT INSERTION | 10061657 |
| MESENTERIC ARTERY STENOSIS | 10027396 |
| THROMBOTIC THROMBOCYTOPENIC PURPURA | 10043648 |
| PERIPHERAL ARTERY ANGIOPLASTY | 10057518 |
| | 10020027 |
| RETINAL ARTERY OCCLUSION | 10038827 |
| RETINAL ARTERY OCCLUSION ARTERIAL THERAPEUTIC PROCEDURE | 10052949 |

**Table 9.11 Arterial** 

| Table 9.11 Afterial | |
|---|---|
| AEDECOD in Upper Case | PT Code |
| ISCHAEMIC STROKE | 10061256 |
| PRECEREBRAL ARTERY OCCLUSION | 10036511 |
| EMBOLIA CUTIS MEDICAMENTOSA | 10058729 |
| EMBOLISM ARTERIAL | 10014513 |
| POST PROCEDURAL MYOCARDIAL INFARCTION | 10066592 |
| RENAL EMBOLISM | 10063544 |
| PERIPHERAL EMBOLISM | 10061340 |
| LERICHE SYNDROME | 10024242 |
| SUBCLAVIAN ARTERY EMBOLISM | 10042332 |
| RENAL ARTERY THROMBOSIS | 10038380 |
| VISUAL ACUITY REDUCED TRANSIENTLY | 10047532 |
| PERIPHERAL ARTERY OCCLUSION | 10057525 |
| PAPILLARY MUSCLE INFARCTION | 10033697 |
| BASILAR ARTERY OCCLUSION | 10048963 |
| PAPILLARY MUSCLE INFARCTION BASILAR ARTERY OCCLUSION BASILAR ARTERY OCCLUSION Ala. For non-commercial use only and all al | |
| Sty of Lakeda. For | |

Table 9.12 Venous

| Tubic 7.12 Tellous | |
|--------------------------------------|----------|
| AEDECOD in Upper Case | PT Code |
| RETINAL VEIN OCCLUSION | 10038907 |
| CEREBRAL VENOUS SINUS THROMBOSIS | 10083037 |
| VENOGRAM ABNORMAL | 10047209 |
| PORTAL VEIN CAVERNOUS TRANSFORMATION | 10073979 |
| PORTAL VEIN OCCLUSION | 10058989 |
| VENOUS OPERATION | 10062175 |
| OBSTETRICAL PULMONARY EMBOLISM | 10029925 |
| BUDD-CHIARI SYNDROME | 10006537 |
| POST THROMBOTIC SYNDROME | 10048591 |
| VENOUS THROMBOSIS | 10047249 |
| PULMONARY THROMBOSIS | 10037437 |
| PULMONARY VEIN OCCLUSION | 10068690 |
| VENOOCCLUSIVE DISEASE | 10062173 |
| VENOUS REPAIR | 10052964 |
| POSTOPERATIVE THROMBOSIS | 10050902 |
| CAVERNOUS SINUS THROMBOSIS | 10007830 |
| VENOUS RECANALISATION | 10068605 |
| HEPATIC VEIN THROMBOSIS | 10019713 |
| THROMBOPHLEBITIS MIGRANS | 10043581 |
| DEEP VEIN THROMBOSIS POSTOPERATIVE | 10066881 |
| MESENTERIC VENOUS OCCLUSION | 10027403 |
| PULMONARY VENO-OCCLUSIVE DISEASE | 10037458 |
| SPLENIC VEIN OCCLUSION | 10068122 |
| EMBOLISM VENOUS | 10014522 |
| TRANSVERSE SINUS THROMBOSIS | 10044457 |
| SI QIII TIII PATTERN | 10068479 |
| SPLENIC VEIN THROMBOSIS | 10041659 |
| VENA CAVA FILTER REMOVAL | 10074397 |
| VENOCCLUSIVE LIVER DISEASE | 10047216 |
| RENAL VEIN THROMBOSIS | 10038548 |
| VENOUS THROMBOSIS NEONATAL | 10064602 |
| POST PROCEDURAL PULMONARY EMBOLISM | 10063909 |
| VENOUS THROMBOSIS IN PREGNANCY | 10067030 |
| ILIAC VEIN OCCLUSION | 10058992 |
| RENAL VEIN EMBOLISM | 10038547 |
| VENOUS THROMBOSIS LIMB | 10061408 |

Table 9.12 Venous

| Table 9.12 Venous | |
|------------------------------------|----------|
| AEDECOD in Upper Case | PT Code |
| THROMBOPHLEBITIS | 10043570 |
| RENAL VEIN OCCLUSION | 10056293 |
| PELVIC VENOUS THROMBOSIS | 10034272 |
| PENILE VEIN THROMBOSIS | 10034324 |
| OVARIAN VEIN THROMBOSIS | 10072059 |
| JUGULAR VEIN OCCLUSION | 10076835 |
| VENA CAVA THROMBOSIS | 10047195 |
| MAHLER SIGN | 10075428 |
| PHLEBECTOMY | 10048874 |
| VENOUS STENT INSERTION | 10063389 |
| PULMONARY MICROEMBOLI | 10037421 |
| SUPERIOR SAGITTAL SINUS THROMBOSIS | 10042567 |
| SUPERIOR VENA CAVA SYNDROME | 10042569 |
| VENA CAVA EMBOLISM | 10047193 |
| INFERIOR VENA CAVAL OCCLUSION | 10058987 |
| JUGULAR VEIN THROMBOSIS | 10023237 |
| PULMONARY EMBOLISM | 10037377 |
| VENA CAVA FILTER INSERTION | 10048932 |
| COMPRESSION GARMENT APPLICATION | 10079209 |
| PULMONARY VENOUS THROMBOSIS | 10037459 |
| CATHETERISATION VENOUS | 10052698 |
| SUPERFICIAL VEIN THROMBOSIS | 10086210 |
| PORTAL VEIN THROMBOSIS | 10036206 |
| POSTPARTUM VENOUS THROMBOSIS | 10036300 |
| HEPATIC VEIN OCCUSION | 10058991 |
| SUPERIOR VENA CAVA OCCLUSION | 10058988 |
| OPHTHALMIC VEIN THROMBOSIS | 10074349 |
| OBSTRUCTIVE SHOCK | 10073708 |
| RETINAL VEIN THROMBOSIS | 10038908 |
| THROMBOPHLEBITIS NEONATAL | 10043586 |
| INFERIOR VENA CAVA SYNDROME | 10070911 |
| THROMBOSIS CORPORA CAVERNOSA | 10067270 |
| PULMONARY INFARCTION | 10037410 |
| SUBCLAVIAN VEIN THROMBOSIS | 10049446 |
| HOMANS' SIGN POSITIVE | 10051031 |
| VENOUS OCCLUSION | 10058990 |
| THROMBOSED VARICOSE VEIN | 10043605 |

Table 9.12 Venous

| AEDECOD in Upper Case | PT Code |
|--------------------------------|----------|
| AXILLARY VEIN THROMBOSIS | 10003880 |
| DEEP VEIN THROMBOSIS | 10051055 |
| PAGET-SCHROETTER SYNDROME | 10050216 |
| MAY-THURNER SYNDROME | 10069727 |
| CEREBRAL VENOUS THROMBOSIS | 10008138 |
| BRACHIOCEPHALIC VEIN OCCLUSION | 10076837 |
| MESENTERIC VEIN THROMBOSIS | 10027402 |
| CENTRAL VENOUS CATHETERISATION | 10053377 |

# Table 9.13 Vessel unspecified/unknown

| AEDECOD in Upper Case | PT Code |
|------------------------------------|----------|
| HEPATIC INFARCTION | 10019680 |
| ARTERIOVENOUS FISTULA OCCLUSION | 10058562 |
| VASCULAR GRAFT OCCLUSION | 10049060 |
| PNEUMATIC COMPRESSION THERAPY | 10059829 |
| ARTERIOVENOUS FISTULA THROMBOSIS | 10003192 |
| TESTICULAR INFARCTION | 10043337 |
| SPLENIC INFARCTION | 10041648 |
| CEREBROSPINAL THROMBOTIC TAMPONADE | 10052173 |
| DEVICE EMBOLISATION | 10074896 |
| PARAPLEGIA | 10033892 |
| CEREBRAL INFARCTION FOETAL | 10008119 |
| TUMOUR EMBOLISM | 10045168 |
| CEREBROVASCUL AR ACCIDENT | 10008190 |
| STOMA SITE THROMBOSIS | 10074515 |
| THROMBECTOMY | 10043530 |
| INTRACARDIAC THROMBUS | 10048620 |
| HEMIPLEGIA | 10019468 |
| CÉRÉBRAL CONGESTION | 10076929 |
| CEREBELLAR INFARCTION | 10008034 |
| PARAPARESIS | 10033885 |
| PLACENTAL INFARCTION | 10064620 |
| PARESIS | 10033985 |
| PERIPHERAL REVASCULARISATION | 10053351 |
| QUADRIPLEGIA | 10037714 |

Table 9.13 Vessel unspecified/unknown

| AEDECOD in Upper Case | PT Code |
|-----------------------------------------|----------|
| THALAMIC INFARCTION | 10064961 |
| GRAFT THROMBOSIS | 10051269 |
| EMBOLISM | 10061169 |
| CARDIAC VENTRICULAR THROMBOSIS | 10053994 |
| INNER EAR INFARCTION | 10070754 |
| PITUITARY INFARCTION | 10035092 |
| VASCULAR STENT THROMBOSIS | 10063934 |
| CORONARY BYPASS THROMBOSIS | 10059025 |
| INSTILLATION SITE THROMBOSIS | 10073625 |
| ULTRASOUND DOPPLER ABNORMAL | 10045413 |
| FOETAL CEREBROVASCULAR DISORDER | 10053601 |
| INCISION SITE VESSEL OCCLUSION | 10076839 |
| ATRIAL THROMBOSIS | 10048632 |
| CEREBRAL THROMBOSIS | 10008132 |
| APPLICATION SITE THROMBOSIS | 10076026 |
| EMBOLIC STROKE | 10014498 |
| ADRENAL THROMBOSIS | 10075178 |
| BRAIN STEM INFARCTION | 10006147 |
| HAEMORRHAGIC CEREBRAL INFARCTION | 10019005 |
| VASCULAR GRAFT THROMBOSIS | 10069922 |
| MEDICAL DEVICE SITE THROMBOSIS | 10076145 |
| MESENTERIC VASCULAR OCCUUSION | 10074583 |
| DIRECTIONAL DOPPLER FLOW TESTS ABNORMAL | 10013048 |
| VACCINATION SITE THROMBOSIS | 10076190 |
| INFUSION SITE THROMBOSIS | 10065489 |
| EMBOLIC CEREBRAL INFARCTION | 10060839 |
| THROMBOSIS | 10043607 |
| CEREBRAL (SCHAEMIA | 10008120 |
| IMPLANT SITE THROMBOSIS | 10063868 |
| HAEMORRHAGIC TRANSFORMATION STROKE | 10055677 |
| MESENTERIC VASCULAR INSUFFICIENCY | 10027401 |
| VASODILATION PROCEDURE | 10058794 |
| POSTPARTUM THROMBOSIS | 10077022 |
| OPTIC NERVE INFARCTION | 10030936 |
| THROMBOTIC STROKE | 10043647 |
| HAEMORRHOIDS THROMBOSED | 10019023 |
| HAEMORRHAGIC INFARCTION | 10019013 |

Table 9.13 Vessel unspecified/unknown

| AEDECOD in Upper Case | PT Code |
|---------------------------------------------------|----------|
| BONE INFARCTION | 10049824 |
| INTRACARDIAC MASS | 10066087 |
| INJECTION SITE THROMBOSIS | 10022104 |
| CEREBRAL INFARCTION | 10008118 |
| VASCULAR GRAFT | 10067740 |
| EMBOLIC PNEUMONIA | 10065680 |
| CEREBROVASCULAR OPERATION | 10051902 |
| CEREBROVASCULAR DISORDER | 10008196 |
| ANGIOGRAM ABNORMAL | 10060956 |
| THYROID INFARCTION | 10043742 |
| MICROEMBOLISM | 10073734 |
| INFARCTION | 10061216 |
| ADMINISTRATION SITE THROMBOSIS | 10075968 |
| VASCULAR STENT OCCLUSION | 10077143 |
| DISSEMINATED INTRAVASCULAR COAGULATION IN NEWBORN | 10013443 |
| HAEMORRHAGIC STROKE | 10019016 |
| VASCULAR STENT INSERTION | 10063382 |
| PROSTHETIC VESSEL IMPLANTATION | 10068628 |
| SPLENIC THROMBOSIS | 10074601 |
| COLLATERAL CIRCULATION | 10069729 |
| QUADRIPARESIS | 10049680 |
| THROMBOSIS MESENTERIC VESSEL | 10043626 |
| THROMBOTIC CEREBRAL INFARCTION | 10067347 |
| UMBILICAL CORD OCCLUSION | 10076714 |
| CEREBELLAR EMBOLISM | 10067167 |
| DEVICE OCCLUSION | 10064685 |
| VESSEL PUNCTURE SITE OCCLUSION | 10076838 |
| MONOPLEGIA | 10027926 |
| HEPATIC VASCULAR THROMBOSIS | 10074494 |
| DISSEMINATED INTRAVASCULAR COAGULATION | 10013442 |
| RETINAL INFARCTION | 10051742 |
| BRAIN STEM STROKE | 10068644 |
| CEREBRAL SEPTIC INFARCT | 10070671 |
| VISUAL MIDLINE SHIFT SYNDROME | 10066856 |
| MONOPARESIS | 10027925 |
| INTESTINAL INFARCTION | 10022657 |
| ULTRASONIC ANGIOGRAM ABNORMAL | 10061604 |

Table 9.13 Vessel unspecified/unknown

| AEDECOD in Upper Case | PT Code |
|--------------------------------------|----------|
| BRAIN STEM EMBOLISM | 10074422 |
| THROMBOLYSIS | 10043568 |
| RENAL VASCULAR THROMBOSIS | 10072226 |
| RETINAL VASCULAR THROMBOSIS | 10062108 |
| THROMBOSIS PROPHYLAXIS | 10043634 |
| SURGICAL VASCULAR SHUNT | 10058408 |
| SHUNT THROMBOSIS | 10059054 |
| RENAL INFARCT | 10038470 |
| PORTAL SHUNT | 10036204 |
| PARADOXICAL EMBOLISM | 10066059 |
| CEREBROVASCULAR ACCIDENT PROPHYLAXIS | 10049165 |
| SPINAL CORD INFARCTION | 10058571 |
| VESSEL PUNCTURE SITE THROMBOSIS | 10070649 |
| ANGIOGRAM PERIPHERAL ABNORMAL | 10057517 |
| CHOROIDAL INFARCTION | 10057403 |
| VASCULAR OPERATION | 10049071 |
| POST PROCEDURAL STROKE | 10066591 |
| THROMBOANGIITIS OBLITERANS | 10043540 |
| HEPARIN-INDUCED THROMBOCYTOPENIA | 10062506 |
| BRAIN STEM THROMBOSIS | 10062573 |
| SHUNT OCCLUSION | 10040621 |
| TUMOUR THROMBOSIS | 10068067 |
| UMBILICAL CORD THROMBOSIS | 10071652 |
| ANGIOGRAM CEREBRAL ABNORMAL | 10052906 |
| THROMBOSIS IN DEVICE | 10062546 |
| DIPLEGIA | 10013033 |
| BASAL GANGLIA STROKE | 10071043 |
| HEMIPARESIS | 10019465 |
| PANCREATIC INFARCTION | 10068239 |

## 9.3 Assignment of R-ODS Centile Metric Scores

Derive the R-ODS score converted to a percentage value for CIDP according to the table below for listing.

**R-ODS Score Conversion** Table 10

| 1 able 10 R-ODS Score Conversion | |
|-----------------------------------------------|---------------------|
| R-ODS Total Score<br>(R-ODS summed raw score) | Centile Metric |
| Value where PARAMCD = | Value where Derived |
| "SIRODS" | PARAMCD = "CRODS" |
| 0 | 0 |
| 1 | 6 |
| 2 | 11 |
| 3 | 14 |
| 4 | 16 |
| 5 | 19 |
| 6 | 21 |
| 7 | 22 |
| 8 | 24 |
| 9 | 26 |
| 10 | 27 |
| 11 | 28 |
| 12 | 30 |
| 13 | 31 |
| 14 | 32 |
| 15 | 34 |
| 16 | 35 |
| 17 | 36 |
| 18 | 37 |
| 19 | 39 |
| 20 | 40 |
| 21 | 41 |
| 22 | 42 |
| 23 | 43 |
| 24 | 45 |
| 25 | 46 |
| 26 | 47 |
| 27 | 48 |
| 28 | 50 |
| 29 | 51 |
| 30 | 52 |
| 31 | 54 |
| 32 | 55 |
| 33 | 57 |
| 34 | 58 |
| 35 | 60 |
| 36 | 61 |
| 37 | 63 |

and subject to the applicable Terms of Use

| TAK-7<br>Statisti | 71-3002<br>cal Analysis Plan v3.0 | | Page 77 of 77<br>17-Oct-2024 |
|---|---|---|---|
| 1 | 38 | <br> 65 | 16 |
| | 39 | 67 | |
| | 40 | 69 | |
| | 41 | 71 | |
| | 42 | 73 | X 8), |
| | 43 | 76 | |
| | 44 | 80 | |
| | 45 | 83 | : Car |
| | 46 | 88 | |
| | 47 | 93 | 26 <sub>k</sub> |
| | 48 | 100 | |
| | | mercial use only | Page 77 of 77 17-Oct-2024 19 For higher. |
| | or non-co | | |